

# **Clinical Study Protocol**

Study Title: An Open-Label, Long-Term Extension Study to Evaluate the Safety and

Efficacy of Tapinarof Cream 1% in Subjects with Atopic Dermatitis

Protocol No.: DMVT-505-3103

Clinical Study Protocol

Sponsor: Dermavant Sciences, Inc.

3300 Paramount Parkway, Suite 150

Morrisville, NC, USA 27560

Compound Name: Tapinarof (DMVT-505)

Protocol Number: DMVT-505-3103

Indication: Atopic Dermatitis

Development Phase: 3

IND Number: 104601

Current Version: 2.0

Original Protocol 4/18/2021

Approved/Effective Date

Amendment 1 6/16/2021

Approved/Effective Date:

### **Confidentiality Statement**

The information contained in this document, particularly unpublished data, is the property or under control of Dermavant Sciences, Inc., and is provided to you in confidence as an investigator, potential investigator, or consultant, for review by you, your staff, and an applicable Institutional Review Board or Independent Ethics Committee. The information is only to be used by you in connection with authorized clinical studies of the investigational drug described in the protocol. You will not disclose any of the information to others without written authorization from Dermavant Sciences, Inc., except to the extent necessary to obtain informed consent from those persons to whom the drug may be administered.

# **Sponsor Signature Page**


Clinical Study Protocol

**Study Title:** An Open-Label, Long-Term Extension Study to Evaluate the Safety and Efficacy of

Tapinarof Cream 1% in Subjects with Atopic Dermatitis

**Protocol Number:** DMVT-505-3103

This protocol has been approved by a representative of Dermavant Sciences, Inc. The following signature documents this approval.



This electronic signature is legally binding equivalent of traditional handwritten signatures and is captured in the audit trail of the document.

# **Medical Monitor / Sponsor Information Page**


Clinical Study Protocol

Medical Monitor/Serious Adverse Event (SAE) Contact Information

| Role | Name | Daytime Phone Number and Email<br>Address | After-hours<br>Phone/Cell/Pager<br>Number |
|---|---|---|---|
| Primary Medical Monitor | | | |
| Secondary Medical Monitor | | | |
| Serious Adverse Event (SAE)/<br>Pregnancy Reporting Contact<br>Information | North America Safety<br>Mailbox | | N/A |

# **Study Sponsor**

This study is sponsored by Dermavant Sciences, Inc.

# **Sponsor Registered Address and Regulatory Contact**

Dermavant Sciences, Inc. 3300 Paramount Parkway, Suite 150 Morrisville, NC 27560 USA

# **Investigator Statement**


Clinical Study Protocol

**Study Title:** An Open-Label, Long-Term Extension Study to Evaluate the Safety and Efficacy of Tapinarof Cream 1% in Subjects with Atopic Dermatitis

- I confirm agreement to conduct the study in compliance with the protocol.
- I acknowledge that I am responsible for overall study conduct. I agree to personally conduct or supervise the described study.
- I agree to ensure that all associates, colleagues, and employees assisting in the conduct of the study are informed about their obligations and comply with the study protocol. Mechanisms are in place to ensure that site staff receives the appropriate information throughout the study.

| Principal Investigator Name | Signature |
|-----------------------------|-----------|
| - | - |
| Date | Site |

# **Table of Contents**

| Synopsis | | 12 |
|---|---|---|
| 1 | Introduction | 23 |
| 1.1 | Background Information and Study Rationale | 23 |
| 1.1.1 | Background Information | |
| 1.1.2 | Study Rationale | 24 |
| 1.2 | Rationale for Study Design, Dose, and Control Groups | 25 |
| 1.3 | Potential Risks and Benefits | 25 |
| 1.3.2 | Benefit Assessment. | 26 |
| 1.3.3 | Overall Benefit Risk | 26 |
| 2 | Objectives and Endpoints | 27 |
| 3 | Study Design. | 29 |
| 3.1 | Overall Design | 29 |
| 3.2 | Treatment Groups and Duration | 30 |
| 4 | Study Population | 31 |
| 4.1 | Type and Number of Subjects | 31 |
| 4.2 | Inclusion Criteria | 31 |
| 4.3 | Exclusion Criteria | 32 |
| 4.4 | Lifestyle Restrictions | 35 |
| 4.5 | Withdrawal Criteria | 35 |
| 4.5.1 | Reasons for Withdrawal from the Study | 35 |
| 4.5.2 | Withdrawal Procedures | 36 |
| 4.6 | Lost to Follow-Up | 36 |
| 5 | Study Treatment | 37 |
| 5.1 | Study Drug | 37 |
| 5.1.1 | Description, Packaging, and Labeling | 37 |
| 5.1.2 | Storage | 37 |
| 5.1.3 | Handling and Disposal | 37 |
| 5.1.4 | Preparation | 37 |
| 5.1.5 | Administration of Study Drug | 37 |
| 5.1.5.1 | Treatment Based on Validated Investigator Global Assessment of Atopic Dermatitis | 37 |

| 5.1.5.2 | Disease Worsening (Validated Investigator Global Assessment of Atopic Dermatitis ≥ 2 During the Study) | 38 |
|---|---|---|
| 5.1.5.3 | Application of Study Drug | 38 |
| | | 39 |
| 5.2 | Randomization/Treatment Assignment | 39 |
| 5.3 | Blinding | 40 |
| 5.4 | Compliance with Study Drug Administration | 40 |
| 5.5 | Treatment after the End of the Study | 40 |
| 5.6 | Prior and Concomitant Therapy | 40 |
| 5.6.1 | Permitted Medications and Nondrug Therapies | 41 |
| 5.6.2 | Prohibited Medications and Nondrug Therapies | 41 |
| 6 | Study Assessments and Procedures | 43 |
| 6.1 | Medical History, Demography, and Baseline Characteristics | 43 |
| 6.1.1 | Demographics | 43 |
| 6.1.2 | Medical History | 43 |
| 6.2 | Safety Assessments | 43 |
| 6.2.1 | Adverse Events | 43 |
| 6.2.2 | Brief Physical Examination | 43 |
| 6.2.3 | Vital Signs | 44 |
| 6.2.4 | Clinical Safety Laboratory Assessments | 44 |
| 6.2.5 | | 45 |
| 6.2.5.1 | | 45 |
| 6.2.5.2 | | 45 |
| 6.3 | Efficacy Assessments | 46 |
| 6.3.1 | Assessments Completed by Investigator | 46 |
| 6.3.1.1 | Validated Investigator Global Assessment of Atopic Dermatitis | 46 |
| 6.3.1.2 | Body Surface Area Affected. | 46 |
| 6.3.1.3 | Eczema Area and Severity Index | 46 |
| 6.3.2 | Assessments Completed by Subject or Caregiver | 47 |
| 6.3.2.1 | | 47 |
| 6.3.2.2 | | 47 |
| 6.3.2.3 | Peak Pruritus-Numeric Rating Scale | 47 |
| 6.3.2.4 | | 48 |
| 6.3.2.5 | | 48 |
| 6.3.2.6 | | 49 |

| Derma vant s | Sciences, inc. | innear Study 1 Totocc |
|---|---|---|
| 6.3.3 | Optional Clinical Photography | 49 |
| 6.4 | Treatment of Study Drug Overdose | 49 |
| 6.5 | Virtual Assessments | 49 |
| 7 | Timing of Procedures and Assessments | 51 |
| 7.1 | Visit 0; Screening Period for Direct-Enrolling Subjects (Day -30 to Day -1) | 51 |
| 7.2 | Visit 1; Baseline (Day 1) | 51 |
| 7.2.1 | Baseline Visit for Subjects Rolling Over from DMVT-505-3101 and DMVT-50 | 5-310251 |
| 7.2.2 | Baseline Visit for Subjects Rolling Over from DMVT-505-2104 | 52 |
| 7.2.3 | Baseline Visit for Subjects Enrolling Directly into DMVT-505-3103 | 53 |
| 7.3 | Visits 2 to 13; Treatment Period | 54 |
| 7.4 | Phone Contact at Week 2 (Day 15 ± 3 Days) | 55 |
| 7.5 | Follow-Up Visit 14; Week 49 (Day 344 ±3 Days) | 55 |
| 7.6 | Unscheduled Visits | 56 |
| 7.7 | Early Termination Visit | 56 |
| 7.8 | End of Study | 57 |
| 8 | Safety Monitoring and Reporting | 58 |
| 8.1 | Adverse Events, Serious Adverse Events, and Adverse Events of Special Interes | t58 |
| 8.1.1 | Definition of Adverse Events | 58 |
| 8.1.2 | Definition of Serious Adverse Event | 59 |
| 8.1.3 | Adverse Events of Special Interest | 60 |
| 8.2 | Classification of Adverse Events | 61 |
| 8.2.1 | Assigning Severity Rating for Adverse Events | 61 |
| 8.2.1.1 | Criteria for Determining Adverse Event Severity | 61 |
| 8.2.1.2 | Toxicity Management Criteria | 61 |
| 8.2.1.2.1 | Grade 1 or Grade 2 Adverse Event | 61 |
| 8.2.1.2.2 | Grade 3 Adverse Event | 61 |
| 8.2.1.2.3 | Grade 4 Adverse Event | 61 |
| 8.2.1.2.4 | Folliculitis | 62 |
| 8.2.1.2.5 | Other Management Criteria: | 62 |
| 8.2.2 | Assigning Causal Relationship to Study Drug | 62 |
| 8.3 | Time Period and Frequency for Event Assessment and Follow-Up | 62 |
| 8.3.1 | Adverse Event Reporting | 62 |
| 8.3.2 | Follow-Up of Adverse Events | 63 |
| 8.4 | Reporting Procedures | 63 |
| 8.4.1 | Serious Adverse Event Reporting | 63 |

| 8.4.2 | Regulatory Reporting Requirements for Serious Adverse Events | 63 |
|---|---|---|
| 8.5 | Pregnancy Management and Reporting | 64 |
| 9 | Data Management | |
| 10 | Statistical Considerations and Data Analyses | 66 |
| 10.1 | General Considerations | 66 |
| 10.2 | Determination of Sample Size | 66 |
| 10.3 | Analysis Populations | 66 |
| 10.4 | Planned Analyses | 66 |
| 10.4.1 | Disposition and Demographics | 66 |
| 10.4.2 | Efficacy Analyses | 66 |
| 10.4.3 | Safety Analyses | 68 |
| 10.4.4 | | 68 |
| 10.4.5 | | 69 |
| 10.5 | Interim Analyses | 69 |
| 10.6 | Handling of Missing Data | 69 |
| 11 | Responsibilities | 70 |
| 11.1 | Investigator Responsibilities | 70 |
| 11.1.1 | Good Clinical Practice | 70 |
| 11.1.2 | Institutional Review Board/Independent Ethics Committee Approval | 70 |
| 11.1.3 | Informed Consent/Assent | 70 |
| 11.1.4 | Confidentiality | 70 |
| 11.1.5 | Study Files and Retention of Records | 71 |
| 11.1.6 | Electronic Case Report Forms | 72 |
| 11.1.7 | Drug Accountability | |
| 11.1.8 | Inspections | 72 |
| 11.1.9 | Protocol Compliance | 72 |
| 11.2 | Sponsor Responsibilities | 73 |
| 11.2.1 | Protocol Modifications | 73 |
| 11.2.2 | Study Report and Publications | 73 |
| 11.2.3 | Posting of Information on Publicly Available Clinical Trial Registers | 73 |
| 11.3 | Joint Investigator/Sponsor Responsibilities | 73 |
| 11.3.1 | Access to Information for Monitoring | 73 |
| 11.3.2 | Access to Information for Auditing or Inspections | 74 |
| 11.3.3 | Study Discontinuation | 74 |
| 12 | References | 75 |

Confidential Page | 9

Table 6:

Table 7: Table 8: National Cancer Institute CTCAE 61

# **Table of Abbreviations**

| Term | Full Description |
|-----------|------------------------------------------------------|
| AD | atopic dermatitis |
| AE | adverse event |
| AESI | adverse event of special interest |
| AhR | Aryl hydrocarbon receptor |
| ALT | alanine aminotransferase |
| Anti-HBc | anti-hepatitis B core antigen |
| Anti-HBs | anti-hepatitis B surface antigen |
| ARNT | AhR nuclear translocator |
| AST | aspartate aminotransferase |
| BID | twice daily |
| BMI | body mass index |
| BSA | body surface area |
| %BSA | percent of total body surface area |
| BUN | blood urea nitrogen |
| BWTP | Beijing Wenfeng Tianji Pharmaceutical Technology Co. |
| С | collect |
| CFR | Code of Federal Regulations |
| CRF | case report form |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CV | cardiovascular |
| D | dispense |
| Dermavant | Dermavant Sciences, Inc. |
| EASI | Eczema Area and Severity Index |
| ET | early termination |
| FU | follow-up |
| GSK | GlaxoSmithKline |
| HBsAg | hepatitis B surface antigen |
| ICF | informed consent form |
| ICH | International Council for Harmonisation |
| IEC | Independent Ethics Committee |
| IL | interleukin |
| IRB | Institutional Review Board |
| ITT | Intent-to-Treat |
| JAK | Janus kinase |
| LOCF | last observation carried forward |
| MCH | mean corpuscular hemoglobin |
| MCHC | mean corpuscular hemoglobin concentration |
| MCV | mean corpuscular volume |
| NA | not applicable |
| Nrf2 | nuclear factor erythroid 2-related factor 2 |
| OC | observed case |
| OL-LTE | open-label, long-term extension |

| Dermayant Sciences | s, inc. Clinical Study Protoco |
|---|---|
| Term | Full Description |
| P/C | phone contact |
| PGA | Physician's Global Assessment |
| PK | pharmacokinetic(s) |
| PP-NRS | Peak Pruritus-Numeric Rating Scale |
| QD | once daily |
| RBC | red blood cell(s) |
| SAE | serious adverse event |
| SD | standard deviation |
| TAMA | therapeutic AhR-modulating agent |
| TEAE | treatment-emergent adverse event |
| ULN | upper limit of normal |
| US | United States |
| V | visit |
| vIGA-AD <sup>TM</sup> | validated Investigator Global Assessment for Atopic Dermatitis |
| WBC | white blood cell(s) |
| WOCBP | women of child-bearing potential |

**Tapinarof** Protocol No.: DMVT-505-3103 Dermavant Sciences, Inc. Clinical Study Protocol

### **Synopsis**

| Name of Sponsor/Co | ompany: | | | | |
|---|---|---|---|---|---|
| Dermavant Sciences, | Inc. | | | | |
| Name of Investigation | onal Product: | | | | |
| DMVT-505 (tapinaro | of cream, 1%) | | | | |
| Name of Active Ingi | redient: | | | | |
| Tapinarof | | | | | |
| <b>Protocol Number:</b> | DMVT-505-3103 | Phase: | 3 | Country: | United States (US) and Canada |
| Title of Study: | | | | <u>.</u> | • |

An Open-Label, Long-Term Extension Study to Evaluate the Safety and Efficacy of Tapinarof Cream 1% in Subjects with Atopic Dermatitis

#### **Study Site(s):**

Up to approximately 135 sites in the US and Canada

### **Objectives:**

- To evaluate the safety and tolerability of tapinar fcream, 1% in subjects with atopic dermatitis (AD)
- To evaluate the efficacy of tapinar f cream, 1% over an extended period of time in subjects with AD
- To describe the effect of tapinar f cream, 1% on AD symptom severity and the associated impact on daily activities and attitudes in subjects with AD

# Methodology:

This is an open-label, long-term multicenter, study to evaluate the safety and efficacy of topical tapinarof cream, 1% in subjects with AD. Subjects in this study will have either: a) completed treatment with tapinarof or vehicle in one of two Phase 3 pivotal safety and efficacy studies, DMVT-505-3101 or DMVT-505-3102, and rolled over into this study; b) completed treatment with tapinarof in the Phase 2 maximal use pharmacokinetics [PK] study, DMVT-505-2104, and rolled over into this study; or c) enrolled directly into this study. This study will consist of up to 48 weeks of treatment and a 1-week safety follow-up period. At the completion of the Week 8 visit of study DMVT-505-3101 or study DMVT-505-3102 or the Day 28 visit of study DMVT-505-2104 (Baseline [Day 1] in this study), all eligible subjects will be offered enrollment in this open-label long-term extension (OL-LTE) study. Approximately 125 additional pediatric subjects ages 2 to < 18 years who are not eligible for participation in the Phase 3 pivotal studies (DMVT-505-3101 or DMVT-505-3102) will be enrolled directly into this OL-LTE study. Study visits during the treatment period for all subjects will occur every 4 weeks (± 3 days). Unscheduled visits may occur, as needed. Subjects who withdraw from the study before Week 48 will return to the study site for an Early Termination visit. The total duration of subject participation in this study will be approximately 49 weeks for rollover subjects (Baseline to Follow-Up) and approximately 53 weeks for direct-enrolling subjects (Screening to Follow-Up).

Rollover subjects in this study will begin treatment based on their validated Investigator Global Assessment in Atopic Dermatitis (vIGA-AD<sup>TM</sup>) score from the final visit in one of the three aforementioned studies (DMVT-505-3101, DMVT-505-3102, or DMVT-505-2104). Subjects entering with a vIGA-AD<sup>TM</sup>  $\geq$  1 will receive treatment once daily (QD) with tapinarof cream, 1% until they achieve a vIGA-AD<sup>TM</sup> score of 0, at which time treatment will be discontinued and subjects monitored for maintenance of disease control (i.e., the extent of the remittive effect). If/when disease worsening occurs, as evidenced by a flare to vIGA-AD<sup>TM</sup> ≥ 2, treatment will be re-initiated and continued until a vIGA-AD<sup>TM</sup> of 0 is achieved. Subjects entering with a vIGA-AD<sup>TM</sup> of 0 will have treatment discontinued beginning at the Baseline visit and will be monitored for maintenance of the remittive effect. If/when disease worsening occurs, as evidenced by a flare to vIGA-AD<sup>TM</sup>  $\geq$  2, treatment will be re-initiated and continued until a vIGA-ADTM of 0 is achieved. This regimen of treatment and re-treatment will continue until the end of the study (i.e., subjects may receive study drug up until the Week 48 visit).

Subjects enrolling directly into this study will receive treatment QD with tapinarof cream, 1% beginning at Baseline and continue treatment until they achieve a vIGA-AD<sup>TM</sup> score of 0, at which time treatment will be discontinued and subjects monitored for maintenance of the remittive effect. If/when disease worsening occurs, as evidenced by a flare to vIGA-AD<sup>TM</sup>  $\geq$  2, treatment will be re-initiated and continued until a vIGA-AD<sup>TM</sup> of 0 is achieved. This regimen of treatment and re-treatment will continue until the end of the study (i.e., subjects may receive study drug up until the Week 48 visit).

Study drug will be dispensed to subjects or their caregivers, applied during the clinic visits, and applied at home between clinic visits as instructed by site personnel. Subjects or their caregivers will be instructed to apply study drug QD to all affected areas, including newly appearing lesions and lesions/areas that improve during the study until a vIGA-AD<sup>TM</sup> of 0 is achieved. Once a vIGA-AD<sup>TM</sup> of 0 is achieved, the treatment period ends. If/when disease worsening occurs, and treatment is re-initiated at a vIGA-AD<sup>TM</sup> of  $\geq 2$ , all lesions currently present and any new lesions that occur during the new treatment period should be treated. Subjects or caregivers will apply sufficient study drug to cover each lesion completely with a thin layer of study drug and will record the time of study drug application and daily itch score (Peak Pruritus-Numeric Rating Scale [PP-NRS]) in a daily diary

Tapinarof Protocol No.: DMVT-505-3103
Dermavant Sciences, Inc. Clinical Study Protocol

provided by the study site. Subjects are allowed, but not required, to treat scalp lesions with study drug; however, efficacy analyses will not include assessment of improvement for AD on the scalp. At the first clinic visit, if applicable, subjects and/or caregivers will be instructed to maintain the approximate dosing time for the daily application of study drug. If applicable to the subject, study drug application instructions will be reviewed at subsequent clinic visits. During subsequent clinic visits, after efficacy and safety assessments (except for Local Tolerability Scale [LTS] if applicable) are completed, subjects or caregivers will apply the study drug to the affected areas while under the supervision of site personnel. The time of the study drug application and assessments will depend on the time of the clinic visit (either morning or afternoon visit). For subjects receiving study drug, subjects should resume their regular chosen application time the following day and thereafter.

### Number of Subjects:

Up to 961 subjects ages 2 years and above will be enrolled in the study, including up to 836 rollover subjects from studies DMVT-505-3101, DMVT-505-3102, and DMVT-505-2104 and approximately 125 subjects enrolling directly into this study.

### Diagnosis and Main Criteria for Inclusion:

### Inclusion Criteria:

Each subject must meet all the following criteria to be eligible to participate in the study:

#### For Rollover Subjects Only:

- 1. Met the criteria as a Study Completer in one of three parent studies (Phase 3 pivotal safety and efficacy study DMVT-505-3101, Phase 3 pivotal safety and efficacy study DMVT-505-3102, or Phase 2 maximal use PK study DMVT-505-2104) and was still receiving study drug at the last visit of one of these studies.
  - NOTE: To meet the criteria as a Study Completer in one of the three parent studies, a subject must have completed  $\geq$  80% of the intended doses in that study.
- 2. Female subjects of childbearing potential must have a negative urine pregnancy test at Baseline (Day 1).

### For Direct-Enrolling Subjects Only:

- 3. Male and female subjects ages 2 years to < 18 years at the time of consent with clinical diagnosis of AD by Hanifin and Rajka criteria.
- 4. Subjects with a vIGA-AD™ score of ≥ 3 and AD covering ≥ 40% of the body surface area (BSA) at Screening and Baseline (pre-randomization), or subjects with a vIGA-AD™ score of 2 at Screening and Baseline (pre-randomization) regardless of BSA. Scalp should be excluded from the BSA calculation to determine eligibility during Screening and at Baseline, and for all efficacy assessments. Subjects must have screened for the DMVT-505-3101 or DMVT-505-3102 study and failed to meet BSA and/or vIGA-AD™ eligibility criteria.
  - NOTE: Subjects with disease only on palms and soles are not eligible.
- 5. AD present for at least 6 months for ages 6 years old and above or 3 months for ages 2 to 5 years old, confirmed by prior medical documentation and/or according to the subject/caregiver report.
- 6. Female subjects of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test at Baseline (Day 1).

#### For All Subjects (Rollover Subjects and Direct-Enrolling Subjects):

- 7. Female subjects of childbearing potential who are engaging in sexual activity that could lead to pregnancy should use one of the following acceptable birth control methods while on study and for 4 weeks after the last exposure to study drug.
  - Acceptable contraception methods include intrauterine device, hormonal contraceptives, barrier method (e.g., condom or diaphragm), or surgical sterilization of male partner (vasectomy)
  - Subjects who claim abstinence as their method of contraception are allowed provided they agree to use a barrier method (e.g., condom or diaphragm) should they become sexually active from Baseline to 4 weeks after the last dose of study drug

Non-child-bearing potential is defined as:

- premenarchal
- pre-menopausal females with a documented bilateral tubal ligation, bilateral oophorectomy, hysterectomy, or hysteroscopic sterilization

Tapinarof Protocol No.: DMVT-505-3103
Dermavant Sciences, Inc. Clinical Study Protocol

• postmenopausal female with a cessation of menses for at least 12 months without an alternative medical cause; a blood sample with follicle stimulating hormone > 40 mIU/mL is confirmatory in questionable cases

8. Subject, subject's parent(s), or legal representative must be capable of giving written informed consent/assent, which includes compliance with the requirements and restrictions listed in the consent/assent form; written informed consent must be obtained prior to any study related procedures.

### **Exclusion Criteria:**

A subject who meets any of the following criteria will be excluded and considered ineligible for participation in the study:

### For Rollover Subjects Only:

- 1. Subjects who were not receiving study drug at the time of the last visit in the parent study (DMVT-505-3101, DMVT-505-3102, or DMVT-505-2104).
- 2. Used a prohibited concomitant product or procedure to treat AD during the parent study.
- 3. Had a serious adverse event (SAE) that was related to treatment or experienced an adverse event (AE) that led to permanent discontinuation of treatment in the parent study.
- 4. Pregnant females as determined by positive urine human chorionic gonadotropin test at Baseline.

### For Direct-Enrolling Subjects Only:

- 5. Concurrent conditions:
  - a. Immunocompromised (e.g., lymphoma, acquired immunodeficiency syndrome) or medical history of positive human immunodeficiency virus antibody at Screening.
  - b. Chronic or acute systemic infection requiring treatment with antiparasitics or antiprotozoals, within 4 weeks prior to the Baseline visit.
  - c. Chronic or acute systemic bacterial infection requiring treatment with systemic antibiotics within one week prior to the Baseline visit.
  - d. Chronic or acute superficial fungal infection requiring treatment with systemic antifungals within one week prior to the Baseline visit.
  - e. Acute active bacterial, fungal, or viral (herpes simplex, herpes zoster, chicken pox) skin infection within 1 week prior to the Baseline visit; the condition should be completely resolved one week prior to Baseline Visit.
  - f. Significant dermatologic or inflammatory condition other than AD that, in the Investigator's opinion, would make it difficult to interpret data or assessments during the study. For example, subjects with an active skin condition such as Kaposi's varicelliform eruption, scabies, molluscum contagiosum, impetigo, psoriasis, severe acne, connective tissue disorder, or Netherton's syndrome, or any other concurrent active disease.
  - g. Concurrent skin lesions in the treatment area or pruritus due to conditions other than AD that, in the opinion of the Investigator, would either interfere with study evaluations or affect the safety of the subject.
- 6. Screening alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥ 2.0 x the upper limit of normal (ULN).
- 7. Screening total bilirubin > 1.5x ULN; total bilirubin > 1.5x ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%.
- 8. Current or chronic history of liver disease, known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones), presence of hepatitis B surface antigen (HBsAg), or positive hepatitis C antibody test result, or presence of anti-hepatitis B core antigen (anti-HBc). Subjects having a negative HBsAg and a positive anti-HBc may enroll if they have a positive anti-hepatitis B surface antigen demonstrating natural immunity. Subjects with a history of hepatitis C virus infection who were medically cured and have an undetectable viral load are eligible to enroll. Subjects with a history of stable non-alcoholic fatty liver disease without evidence of active inflammation (elevated ALT/AST ≥ 2.0x ULN) or cirrhosis are eligible to enroll.
- 9. Current or a history of cancer within 5 years except for adequately treated skin basal cell carcinoma, cutaneous squamous cell carcinoma or carcinoma in situ of the cervix (surgical excision or electrodessication and curettage).
- 10. Pregnant females as determined by positive serum (Screening) or urine (Baseline) human chorionic gonadotropin test.

- 11. Lactating females.
- 12. Previous known participation in a clinical study with tapinarof (previously known as GSK2894512 and WBI-1001).
- 13. Use of any prohibited medication or procedure within the indicated period before the Baseline visit.

NOTE: Prohibited concomitant medications, therapy, etc. during the defined period are as listed in the bullets below. If a subject requires any of these medications throughout the study period, he/she may be excluded from or discontinued from the study, at the discretion of the Investigator and Medical Monitor.

- a. From 4 months prior to Baseline:
  - o DUPIXENT® (dupilumab) injection.
  - Any monoclonal antibody product that becomes approved for AD during the course of the trial.
- b. From 28 days prior to Baseline:
  - Oral, injectable, and suppository preparations of corticosteroids. Eye drops and nasal preparations are allowed. Inhaled preparations are allowed when used for a stable condition and stable dose for ≥ 28 days before Screening and are continued at the same dose throughout the study.
  - Oral preparations and injections of immunosuppressants (cyclosporine, methotrexate, azathioprine, tacrolimus, Janus kinase [JAK] inhibitors, etc.).
  - Excessive sun exposure, tanning booth, other ultraviolet light source and phototherapy including psoralen and ultraviolet A therapy or is unwilling to minimize natural and artificial sunlight exposure.
  - Treatment with antivirals with the exception of short-term treatment for acute upper respiratory viral infections (i.e., influenza) or viral suppressive therapy for a history of recurrent herpes labialis or genital herpes.
- c. From 14 days prior to Baseline:
  - o EUCRISA® (crisaborole) and any other PDE4 inhibitor.
  - o Tacrolimus ointment and pimecrolimus cream.
  - Topical JAK inhibitors.
  - Topical corticosteroids that are classified as medium or high potency (e.g., fluocinonide, triamcinolone acetonide) or super-high potency (e.g., clobetasol propionate). Eye drops and nasal preparations are allowed.
  - Over the counter or herbal medicines for AD (topical and oral preparations). If subjects are using
    emollients, they may continue to use the same emollient on nonlesional skin during the study.
     Emollients containing salicylic acid are prohibited during the study.
- d. From 7 days prior to Baseline:
  - o Topical corticosteroids that are classified as low potency (e.g., desonide, hydrocortisone).
  - Oral, injectable, or intravenous antibiotics or antifungal medications.
  - Topical doxepin, topical gentamicin, or topical neomycin sulfate.

    NOTE: Oral doxepin is allowed for treatment of depression if subject has been on a stable dose (4 weeks) at Screening.
  - Topical products containing urea, except for the treatment of follicular events.
  - Antihistamines/antiallergics (oral, topical and injections): diphenhydramine, chlorpheniramine maleate, hydroxyzine.
    - NOTE: For direct-enrolling subjects, the following antihistamines are allowed from Screening throughout the treatment period: loratadine, fexofenadine hydrochloride, cetirizine hydrochloride. Subjects are allowed to switch from non-allowed antihistamines to allowed antihistamines during Screening but must be on a stable dose for 7 days prior to Baseline.
- e. The subject has received an investigational product within the following time period prior to the first dosing day in the current study: Minimum of 30 days or 5 half-lives of the investigational product (whichever is longer).

For All Subjects (Rollover Subjects and Direct-Enrolling Subjects):

14. A history of or ongoing serious illness or medical, physical, or psychiatric condition(s) that, in the Investigator's opinion, may interfere with the subject's participation in the study, interpretation of results, safety of the subject or ability to understand and give informed consent.

15. Known hypersensitivity to tapinar of or excipients.

#### Investigational Product, Dosage and Mode of Administration:

Tapinarof cream, 1% is a white to off-white cream containing 1% weight/weight (10 mg/gram) tapinarof, supplied in 30-gram tubes, and is to be administered by the subject or their caregiver QD via topical application of a thin layer to affected areas.

### Reference Therapy, Dosage and Mode of Administration:

Not applicable.

### **Duration of Treatment:**

Subjects enrolling in this study may receive treatment for up to 48 weeks. The duration of treatment is based on the vIGA-AD<sup>TM</sup> score. The end of the study is defined as when the last active subject has completed the Follow-up Visit.

### Criteria for Evaluation:



### Study Endpoints:

- Incidence, frequency, and duration of treatment-emergent AEs and SAEs
- Change from Baseline in laboratory values
- Change from Baseline in vital signs

O Proportion of subjects who achieve vIGA-AD<sup>TM</sup> = 0 at least 1 time during the study

0 For subjects entering the study with a vIGA-AD<sup>TM</sup> score  $\geq 2$ : Proportion of subjects who achieved vIGA-AD<sup>TM</sup> = 0 or 1 at least 1 time during the study The following endpoints will be summarized over subjects in the intent-to-treat (ITT) population: change and percent change from Baseline in %BSA affected by visit (OC and LOCF). 0 O change and percent change from Baseline in EASI score by visit (OC and LOCF) O Proportion of subjects with ≥ 50% improvement in EASI score from Baseline by visit (OC and LOCF) 0 Proportion of subjects with ≥ 75% improvement in EASI score from Baseline by visit (OC and LOCF) 0 Proportion of subjects with ≥ 90% improvement in EASI score from Baseline by visit (OC and LOCF) Mean change in PP-NRS score from Baseline at each study visit Proportion of subjects with a Baseline PP-NRS score ≥ 4 who achieve ≥ 4-point reduction in the PP-NRS from Baseline at each study visit


Clinical Study Protocol

#### Statistical Methods:

This is an OL-LTE study, and the number of subjects enrolling is determined in part by subjects completing treatment in one of three parent studies (Phase 3 pivotal safety and efficacy study DMVT-505-3101, Phase 3 pivotal safety and efficacy study DMVT-505-3102, or Phase 2 maximal use PK study DMVT-505-2104) and in part by the number of subjects that enroll directly into this study. A data cut will be made to assess interim results for safety data at the time 100 pediatric subjects (< 18 years of age) have reached 48 weeks of active study drug treatment, inclusive of active study drug treatment in one of three parent studies.

No statistical comparisons will be performed and all study data will be summarized using descriptive statistics for the ITT population overall and by the following categories: received tapinarof treatment in either DMVT-505-3101 or DMVT-505-3102; received vehicle treatment in either DMVT-505-3101 or DMVT-505-3102; received tapinarof treatment in DMVT-505-2104; and enrolled directly into DMVT-505-3103. Categorical variables will be reported using frequency and percentage (e.g., sex, race). Continuous variables will be reported using number of subjects, mean, standard deviation (SD), median, minimum, and maximum.

Demographics, baseline characteristics, and all safety assessments (including LTS assessments), will be summarized using descriptive statistics. Efficacy, functional outcomes, and quality of life assessments will be summarized by mean, SD, median, minimum, and maximum for continuous data, and frequency counts and percentages for categorical data. Median time to event analyses will use the Kaplan-Meier product limit method (if estimable).

# **Schedule of Assessments**

Table 1: Schedule of Assessments

Screening and Baseline Visits, Based on Route of Entry into Study

| | Subjects Rolling Over<br>From DMVT-505-3101 or<br>DMVT-505-3102 | Subjects Rolling Over<br>From DMVT-505-2104 | Subjects Enrolling<br>DMVT-50 | |
|---|---|---|---|---|
| | Visit 1 | Visit 1 | Visit 0 | Visit 1 |
| Procedures and Assessment | Baseline <sup>a</sup><br>Day 1 | Baseline <sup>b</sup><br>Day 1 | Screening<br>Day -30 to Day -<br>1 | Baseline<br>Day 1 |
| Informed consent | X | X | X | |
| Confirm eligibility | X | X | X | X |
| Demographics/Fitzpatrick skin type | [X <sup>c</sup> ] | [X <sup>c</sup> ] | X | |
| Medical History | [X <sup>d</sup> ] | $[X^d]$ | Xe | $X^{f}$ |
| Brief physical examination | [X] | [X] | Xg | X |
| Vital signs <sup>h</sup> | [X] | [X] | X | X |
| Pregnancy test (WOCBP) | [X] | [X] | Xi | $\mathbf{X}^{\mathbf{j}}$ |
| Blood sample for clinical laboratory tests <sup>k</sup> | [X] | [X] | X | $X^1$ |
| Urinalysis | [X] | [X] | X | $X^{m}$ |
| Investigator Assessed | | | | |
| vIGA-AD <sup>TM</sup> score <sup>n</sup> | [X] | [X] | X | X |
| %BSA affected <sup>n</sup> | [X] | [X] | X | X |
| EASI <sup>n</sup> | [X] | [X] | X | X |
| Completed by subject or caregiver | | | | |
| PP-NRS (pre-dose) <sup>p</sup> | [X] | [X] | | X |
| Photograph of disease area <sup>r</sup> | [X] | | | X |
| Adverse events | X | X | X | X |

Protocol No.: DMVT-505-3103 Dermavant Sciences, Inc. Clinical Study Protocol

| Procedures and Assessment |
|-------------------------------------------------------------|
| Concomitant medication |
| Dispense (D) /collect (C) diary <sup>p</sup> |
| Dispense (D) /collect (C) study drug <sup>s</sup> |
| Review instructions for study drug application <sup>t</sup> |
| Study drug application under supervision <sup>s</sup> |

| Subjects Rolling Over<br>From DMVT-505-3101 or<br>DMVT-505-3102 |
|-----------------------------------------------------------------|
| Visit 1 |
| Baseline <sup>a</sup><br>Day 1 |
| X |
| D |
| D |
| X |
| X |

| ] | Subjects Rolling Over<br>From DMVT-505-2104 |
|---|---------------------------------------------|
| | Visit 1 |
| | Baseline <sup>b</sup><br>Day 1 |
| | X |
| | D |
| | D |
| | X |
| | X |

| Subjects Enrolling Directly Into<br>DMVT-505-3103 | |
|---|---|
| Visit 0 Visit 1 | |
| Screening Day -30 to Day - 1 | Baseline<br>Day 1 |
| X | X |
| | D |
| | D |
| | X |
| | X |

Protocol No.: DMVT-505-3103 Clinical Study Protocol

# All Subsequent Visits, Regardless of Method of Entry into Study

| | Long-term Extension Period for All Subjects | | | | | | | | FU | ET | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | P/Cw | V 2 | V 3 | V 4 | V 5 | V 6 | V 7 | V 8 | V 9 | V 10 | V 11 | V12 | V 13 | V 14 | NA NA |
| | Week | Week | Week | Week | Week | Week | Week | Week | Week | Week | Week | Week | Week | Week | 1121 |
| | 2 | 4 | 8 | 12 | 16 | 20 | 24 | 28 | 32 | 36 | 40 | 44 | 48 | 49 | |
| | 1 | Day 29 | Day 57 | Day 85 | Day113 | Day 141 | | <b>Day 197</b> | | Day 253 | Day 281 | Day 309 | <b>Day 337</b> | Day 344 | NA |
| Procedures and | (±3 | (± 3 | (±3 | (±3 | (±3 | (±3 | (±3 | (±3 | (±3 | (±3 | (±3 | (±3 | (±3 | (±3 | |
| Assessment | days) | days) | days) | days) | days) | days) | days) | days) | days) | days) | days) | days) | days) | days) | |
| Brief physical examination | | | | X | | | X | | | X | | | X | X | X |
| Vital signs <sup>h</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Urine pregnancy test<br>(WOCBP) | | X | X | X | X | X | X | X | X | X | X | X | X | | X |
| Blood sample for clinical laboratory tests <sup>k</sup> | | | | X | | | X | | | X | | | X | X | X |
| Urinalysis | | | | | | | | | | | | | X | X | X |
| Investigator Assessed | | | | | | | | | | | | | | | |
| vIGA-AD <sup>TM</sup> score <sup>n</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| %BSA affected <sup>n</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| EASI <sup>n</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Completed by subject or caregiver | | | | | | | | | | | | | | | |
| PP-NRS (pre-dose) p | | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Photograph of disease arear | | | | X | | | X | | | X | | | X | | |

Protocol No.: DMVT-505-3103 Clinical Study Protocol

| | | Long-term Extension Period for All Subjects | | | | | | | | | FU | ETv | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | P/Cw | V 2 | V 3 | V 4 | V 5 | V 6 | V 7 | V 8 | V 9 | V 10 | V 11 | V12 | V 13 | V 14 | NA |
| | Week | Week | Week | Week | Week | Week | Week | Week | Week | Week | Week | Week | Week | Week | |
| | 2 | 4 | 8 | 12 | 16 | 20 | 24 | 28 | 32 | 36 | 40 | 44 | 48 | 49 | |
| | Day 15 | _ | | Day 85 | Day113 | <b>Day 141</b> | <b>Day 169</b> | Day 197 | Day 225 | Day 253 | Day 281 | Day 309 | <b>Day 337</b> | <b>Day 344</b> | NA |
| Procedures and | (±3 | (± 3 | (±3 | (±3 | (±3 | (±3 | (±3 | (±3 | (±3 | (±3 | (±3 | (±3 | (±3 | (±3 | |
| Assessment | days) | days) | days) | days) | days) | days) | days) | days) | days) | days) | days) | days) | days) | days) | |
| Adverse events | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant medication | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Dispense (D) /collect (C) diary <sup>p</sup> | | C/D | C/D | C/D | C/D | C/D | C/D | C/D | C/D | C/D | C/D | C/D | С | | С |
| Review diaries for treatment compliance | | X | X | X | X | X | X | X | X | X | X | X | X | | X |
| Dispense (D) /collect (C) study drug <sup>s</sup> | | C/D | C/D | C/D | C/D | C/D | C/D | C/D | C/D | C/D | C/D | C/D | С | | С |
| Review instructions for study drug application <sup>t</sup> | X | X | X | X | X | X | X | X | X | X | X | X | | | |
| Study drug application under supervision <sup>u</sup> | | X | X | X | X | X | X | X | X | X | X | X | | | |

- a. Baseline Visit to occur at the time of completion of Visit 6 (Week 8) from the DMVT-505-3101 or DMVT-505-3102 studies. Assessments with an unbracketed X should be completed at the Baseline visit. For assessments with a bracketed X, the assessment completed at the final visit of the parent study will be used as the Baseline value for this study.
- b. Baseline Visit to occur at the time of completion of Visit 4 (Day 28) from the DMVT-505-2104 study. Assessments with an unbracketed X should be completed at the Baseline visit. For assessments with a bracketed X, the assessment completed at the final visit of the parent study will be used as the Baseline value for this study.
- c. Demographics/Fitzpatrick skin type as collected at Screening in one of three parent studies (Phase 3 pivotal safety and efficacy study DMVT-505-3101, Phase 3 pivotal safety and efficacy study DMVT-505-3102, or Phase 2 maximal use PK study DMVT-505-2104).
- d. Review medical history as collected in one of three parent studies.
- e. Medical history will include year of AD diagnosis, CV family history, allergic conditions, and risk factors (including height, weight, medical conditions) and family history of liver disease. As part of the subject's medical history, all systemic (oral and injectable) medications used by the subject for treatment of AD prior to 30 days before the Screening visit will be collected.
- f. Review medical history at Baseline and record any changes.
- g. Physical examination will include height and weight (BMI will be calculated in the CRF) at the Screening visit; a brief physical examination will be performed at other visits.
- h. Vital signs will include blood pressure, pulse rate, and body temperature and should be measured after the subject is seated for at least 5 minutes. Vital signs will be measured before blood collection for clinical laboratory assessments (where applicable).
- i. Serum pregnancy test to be performed at the Screening visit only and urine pregnancy test to be performed at subsequent clinic visits when pregnancy testing is performed.
- j. Urine pregnancy test to be performed before randomization.
- k. Includes serum chemistry and liver chemistry tests, and hematology.
- l. Blood sample collection for clinical laboratory tests is not required at the Baseline Visit if it has been  $\leq$ 14 days since samples were collected at Screening and the results of those clinical laboratory tests were within the normal range.
- m. Urine sample collection for urinalysis is not required at the Baseline Visit if it has been  $\leq$ 14 days since samples were collected at Screening and the results of those clinical laboratory tests were within the normal range.

n. The vIGA-AD<sup>TM</sup> assessment should be performed before the %BSA and EASI assessments. The subject's scalp should be excluded from the vIGA-AD<sup>TM</sup>, %BSA, and EASI

calculations. p. Subjects (or caregivers) should perform the PP-NRS assessment daily and record the results in their diary. When subjects apply study drug in the clinic, subjects will not complete the diary at home; application time and PP-NRS will be recorded in the clinic. PP-NRS should be completed every day, even if subjects are not actively applying study drug.

- r. Photography will be performed in a subgroup of subjects at selected study sites. Informed consent/assent and photographic release will be required.
- s. Subjects will be monitored for disease worsening (vIGA-AD<sup>TM</sup>  $\geq$ 2), and study drug may be started at any time during the observation period. If an unscheduled visit is required for re-start of study drug, then the vIGA-AD<sup>TM</sup> must be completed.
- t. For subjects receiving study drug, subjects or their caregivers will be instructed to apply study drug OD at the approximate same time each day, based on subject or caregiver preference.
- u. For subjects receiving study drug, study drug will be applied after safety assessments have been conducted,
- v. Subjects who withdraw from the study before Visit 13 (Week 48) will complete an ET visit. A follow-up visit is not required for a subject who early terminates.
- w. Phone calls to assess AEs and concomitant medications, to review study drug application procedures (if applicable), and to confirm subject's continued participation in the study. Subjects should be reminded to complete the diary and bring it with them to the next clinic visit.
- AD = atopic dermatitis; AE = adverse event (s); BMI = body mass index; %BSA = percent body surface area; C = collect;

; ET = early termination; EASI = Eczema Area and

= case report form; CV = cardiovascular; D = dispense;

 $\frac{1}{2}$ ; NA = not applicable; P/C = phone call; PK = pharmacokinetic;

Severity Index; FU = follow-up;

; PP-NRS = Peak Pruritus-Numeric Rating Scale; QD = once daily; WOCBP = women of child-bearing potential; V = visit; vIGA-AD<sup>1M</sup> = Validated Investigator Global Assessment in Atopic Dermatitis.

### 1 Introduction

# 1.1 Background Information and Study Rationale

# 1.1.1 Background Information

Atopic dermatitis (AD) (also called atopic eczema) is an intensely pruritic, chronic, relapsing, inflammatory skin disease [Bieber, 2008]. The characteristic signs and symptoms of AD include sensations of pruritis and burning, xerosis, erythematous papules and plaques, exudation, crusting, and lichenification. Quality of life is affected through sleep deprivation due to the intense and constant itching, as well as the stigma associated with having a visible skin disease [Carroll, 2005; Lewis-Jones, 2006]. Up to 30% of children may be affected by AD at some point, and 2% to 10% of adults have AD [Bieber, 2008]. Currently there is no curative therapy. Stabilizing the disease and reducing the number and severity of flares are the primary goals of treatment. Topical treatments directed at skin inflammation are a key factor in disease management, as is symptomatic relief of itching. Although multiple topical treatment options are available, there still remains a need for a topical treatment that combines a high level of efficacy with an acceptable safety profile that permits application to a large body surface area (BSA) without restrictions on duration of treatment.

Tapinarof (DMVT-505), formerly known as GSK2894512 and WBI-1001, is a fully synthetic naturally identified stilbene that is being developed by Dermavant Sciences, Inc. (Dermavant) as a novel anti-inflammatory agent for the topical treatment of AD and plaque psoriasis. The compound (number WBI-1001) was initially developed by Welichem Biotech Inc. (Welichem; Burnaby, British Columbia, Canada) and then was acquired by GlaxoSmithKline (GSK) on 31 July 2012 for further development in the rest of the world except China. Dermavant acquired the drug from GSK on 20 August 2018 for continued development in all other territories. Development of tapinarof cream in Japan is being jointly pursued with Japan Tobacco Inc. (JT), with a Phase 3 program in PSO and AD scheduled to commence in late 2021. In China, the compound was independently developed by Beijing Wenfeng Tianji Pharmaceutical Technology Co. (BWTP) (Shenzhen Celestial) under the name benvitimod (active ingredient corresponds to tapinarof). BWTP was granted authorization to market benvitimod cream (a different formulation and excipient profile compared to tapinarof cream) as Symbiox® in China in July 2019.

Tapinarof cream, 1% is a white to off-white, oil-in-water emulsion intended for topical application to AD and psoriatic skin lesions, which has a novel mechanism of action. Tapinarof is a nonsteroidal, small molecule therapeutic aryl hydrocarbon receptor (AhR) modulating agent (TAMA), which exerts its therapeutic effects via agonism of AhR, a cytosolic ligand-dependent transcription factor. Upon ligand binding, AhR translocates to the nucleus and dimerizes with AhR nuclear translocator (ARNT) forming an AhR-ARNT heterodimer [Smith, 2017]. The AhR-ARNT heterodimer modulates gene transcription through direct and indirect interaction with DNA. By activation of this AhR signaling pathway, tapinarof has the potential to downregulate the expression of pro-inflammatory cytokines, including interleukin (IL)-4, IL-5, IL-6, IL-13, IL-17A and F, and eotaxin, and upregulate the expression of several skin barrier proteins, including filaggrin, hornerin, and involucrin. In addition, AhR also activates the antioxidative transcription factor nuclear factor-erythroid 2-related factor-2 (Nrf2), upregulating the expression of antioxidative enzymes [Smith, 2017; Furue, 2019]. By targeting AhR, tapinarof has a biological profile that differs from that of currently available products, offering patients a truly novel therapeutic treatment option for plaque psoriasis and AD.

Two Phase 2b, 12-week, randomized, double-blind, vehicle-controlled, 6-arm, parallel group, dose-finding studies with topically applied tapinarof cream were conducted by GSK; 1 study each in subjects with AD or psoriasis. These 2 studies evaluated the safety and efficacy of tapinarof cream (Formulation F) at

2 concentrations (0.5% or 1% weight/weight [w/w]) and 2 application frequencies (once daily [QD] or twice daily [BID]) in 247 adult and adolescent subjects with AD and in 227 adult subjects with plaque psoriasis. In both studies, tapinarof showed a clear therapeutic effect compared with vehicle, with the 1% w/w concentration treatment groups demonstrating a higher proportion of subjects with treatment success compared with the 0.5% w/w concentration groups (applied QD and BID in the AD study). In both indications, the tapinarof 1% dosing groups showed a faster onset of action than the 0.5% dosing groups, and QD application had similar efficacy to BID application. In both Phase 2b studies, tapinarof showed an acceptable safety profile. Treatment-emergent adverse events (TEAEs) were reported with a higher frequency in the tapinarof groups than in the vehicle groups. The most frequent TEAEs (≥ 5% in any arm or in total) were nasopharyngitis, folliculitis, dermatitis contact, atopic dermatitis, upper respiratory tract infection, headache, vomiting, acne, application site dermatitis, miliaria, dermatitis allergic, and impetigo. The majority of TEAEs were mild or moderate in severity. In each study, the tapinarof 1% QD treatment group had a lower frequency of TEAEs than the tapinarof 1% BID treatment group.


Clinical Study Protocol

Tapinarof has been evaluated in two identical Phase 3, 12-week, randomized, double-blind, vehicle-controlled trials in adult subjects with plaque psoriasis. These studies evaluated the safety and efficacy of tapinarof cream, 1% QD versus vehicle cream QD in a combined 1025 subjects randomized 2:1 tapinarof to vehicle. In both trials, tapinarof demonstrated superiority against vehicle on the primary endpoint, a Physician Global Assessment (PGA) score of 0 (clear) or 1 (almost clear) with a 2-point improvement at Week 12. In addition, tapinarof was highly statistically significant compared to vehicle on all secondary endpoints which included proportion of subjects achieving a 75% improvement in the Psoriasis Area and Severity Index, a PGA score of 0 or 1, change in percent body surface area (%BSA), and proportion of subjects achieving a 90% improvement in the Psoriasis Area and Severity Index at Week 12. TEAEs were reported with a higher frequency in the tapinarof group than in the vehicle group. The most frequent TEAEs (≥ 5% in any arm or in total) were folliculitis, nasopharyngitis, and contact dermatitis. The majority of TEAEs were mild or moderate in intensity.

Tapinarof has also been evaluated in an open-label, long-term extension (OL-LTE) study in adult subjects with plaque psoriasis. The OL-LTE study in adults with plaque psoriasis evaluated the safety and efficacy of tapinarof cream, 1% QD for 40 weeks in 763 subjects enrolled from the two identical 12-week studies. While the study remains ongoing at this time, in a pre-specified interim analysis of the study tapinarof demonstrated continued and substantial improvement in efficacy endpoints beyond the 12 weeks of treatment observed in the identical Phase 3 studies. A high rate of complete disease clearance was achieved, with a remittive effect of approximately 4 months of disease control off therapy. Tapinarof was well tolerated with long-term use and had a safety profile consistent with previous studies.

### 1.1.2 Study Rationale

This 48-week, Phase 3, OL-LTE study is being conducted as part of a clinical development program to evaluate the long-term safety and continued efficacy of tapinarof cream, 1% for the treatment of AD in children and adults. Subjects who complete one of three parent studies (Phase 3 pivotal safety and efficacy study DMVT-505-3101, Phase 3 pivotal safety and efficacy study DMVT-505-3102, or Phase 2 maximal use pharmacokinetics [PK] study DMVT-505-2104) and meet the predefined criteria will have the option to participate in this study. Additionally, approximately 125 pediatric subjects ages 2 to < 18 years who are not eligible for participation in the Phase 3 pivotal studies will also be enrolled directly into this OL-LTE study.

### 1.2 Rationale for Study Design, Dose, and Control Groups

As in the three parent studies, this Phase 3 study will be conducted at multiple study sites in more than one country to enhance the possibility of inclusion of a wider range of population groups and to subsequently increase generalizability of the results. Tapinarof cream is intended for long-term, intermittent use in non-life-threatening inflammatory dermatologic conditions. Therefore, the 48-week duration of long-term, intermittent use of tapinarof cream, 1% in this study is expected to be an adequate duration to assess safety and efficacy of repeated treatment courses of tapinarof as recommended in the International Conference on Harmonisation E1A (ICH E1A) guideline on the extent of population exposure to assess clinical safety for drugs intended for long-term treatment of non-life-threatening conditions, which recommends a minimum of 100 subjects treated with the intended clinical dose to be followed for at least one year.


Clinical Study Protocol

### 1.3 Potential Risks and Benefits

To assess any potential impact on subject eligibility with regard to safety, the Investigator must refer to the current version of the tapinarof Investigator's Brochure for detailed information regarding warnings, precautions, contraindications, adverse events (AEs), and other significant data pertaining to the study drug being used in this study





### 1.3.2 Benefit Assessment

Subjects may experience improvements in their AD during the course of the study and may benefit from the additional safety assessments conducted as part of the study (e.g., physical examination, laboratory tests). Subjects in the study will also contribute to the process of developing a novel anti-inflammatory agent for the topical treatment of AD.

### 1.3.3 Overall Benefit Risk

Taking into account the measures taken to minimize risk to subjects in this study, the potential risks identified in association with tapinarof are justified by the anticipated benefits that may be afforded to subjects with AD.

# 2 Objectives and Endpoints

The objectives and associated endpoints of the study are as follows:

| Objectives | Associated Endpoint |
|---|---|
| To evaluate the safety and tolerability of tapinarof cream, 1% in subjects with AD | <ul> <li>Incidence, frequency, and duration of TEAEs and serious adverse events (SAEs)</li> <li>Change from Baseline in laboratory values</li> <li>Change from Baseline in vital signs</li> </ul> |
| To evaluate the efficacy of tapinarof cream, 1% over an extended period of time in subjects with AD | <ul> <li>For subjects entering the study with a vIGA-AD<sup>TM</sup> score ≥ 1: <ul> <li>Proportion of subjects who achieve vIGA-AD<sup>TM</sup> = 0 at least 1 time during the study</li> <li>For subjects entering the study with a vIGA-AD<sup>TM</sup> score ≥ 2:</li></ul></li></ul> |


Clinical Study Protocol

Protocol No.: DMVT-505-3103 Clinical Study Protocol

| 0 | change and percent change from Baseline in %BSA affected by visit (OC and LOCF) |
|---|---|
| 0 | |
| 0 | change and percent change from Baseline in Eczema Area and Severity Index (EASI) score by visit (OC and LOCF) |
| 0 | Proportion of subjects with ≥ 50% improvement in EASI score from Baseline by visit (OC and LOCF) |
| 0 | Proportion of subjects with ≥ 75% improvement in EASI score from Baseline by visit (OC and LOCF) |
| 0 | Proportion of subjects with $\geq$ 90% improvement in EASI score from Baseline by visit (OC and LOCF) |
| Baseline at 6 • Proportion of | e in Peak Pruritus-Numeric Rating Scale (PP-NRS) score from each study visit of subjects with a Baseline PP-NRS score ≥ 4 who achieve ≥ 4-point the PP-NRS from Baseline at each study visit |
| | Mean chang Baseline at 6 Proportion or reduction in |

### 3 Study Design

# 3.1 Overall Design

This is an open-label, long-term multicenter, study to evaluate the safety and efficacy of topical tapinarof cream, 1% in subjects with AD. Subjects in this study will have either: a) completed treatment with tapinarof or vehicle in one of two Phase 3 pivotal safety and efficacy studies, DMVT-505-3101 or DMVT-505-3102, and rolled over into this study; b) completed treatment with tapinarof in the Phase 2 maximal use PK study, DMVT-505-2104, and rolled over into this study; or c) enrolled directly into this study. This study will consist of up to 48 weeks of treatment and a 1-week safety follow-up period.


Clinical Study Protocol

At the completion of the Week 8 visit of study DMVT-505-3101 or study DMVT-505-3102 or the Day 28 visit of study DMVT-505-2104 (Baseline [Day 1] in this study), all eligible subjects will be offered enrollment in this OL-LTE study. Approximately 125 additional pediatric subjects ages 2 to < 18 years who are not eligible for participation in the Phase 3 pivotal studies (DMVT-505-3101 or DMVT-505-3102) will be enrolled directly into this OL-LTE study. Study visits during the treatment period for all subjects will occur every 4 weeks (± 3 days). Unscheduled visits may occur, as needed. Subjects who withdraw from the study before Week 48 will return to the study site for an Early Termination visit. The total duration of subject participation in this study will be approximately 49 weeks for rollover subjects (Baseline to Follow-Up) and approximately 53 weeks for direct-enrolling subjects (Screening to Follow-Up).

Rollover subjects in this study will begin treatment based on their vIGA-AD<sup>TM</sup> score from the final visit in one of the three aforementioned studies (DMVT-505-3101, DMVT-505-3102, or DMVT-505-2104). Subjects entering with a vIGA-AD<sup>TM</sup>  $\geq$  1 will receive treatment with tapinarof cream, 1% QD until they achieve a vIGA-AD<sup>TM</sup> score of 0, at which time treatment will be discontinued and subjects monitored for maintenance of disease control (i.e., the extent of the remittive effect). If/when disease worsening occurs, as evidenced by a flare to vIGA-AD<sup>TM</sup>  $\geq$  2, treatment will then be re-initiated and continued until a vIGA-AD<sup>TM</sup> of 0 is achieved. Subjects entering with a vIGA-AD<sup>TM</sup> of 0 will have treatment discontinued beginning at the Baseline visit and will be monitored for maintenance of the remittive effect. If/when disease worsening occurs, as evidenced by a vIGA-AD<sup>TM</sup>  $\geq$  2, treatment will then be re-initiated and continued until a vIGA-AD<sup>TM</sup> of 0 is achieved. This treatment and re-treatment pattern of use will be continued until the end of the study (i.e., subjects may receive study treatment up until the Week 48 visit) (see Section 5.1.5.2 for additional details).

Subjects enrolling directly into this study will receive treatment QD with tapinar of cream, 1% beginning at Baseline and continue treatment until they achieve a vIGA-AD<sup>TM</sup> score of 0, at which time treatment will be discontinued and subjects monitored for maintenance of the remittive effect. If/when disease worsening occurs, as evidenced by a flare to vIGA-AD<sup>TM</sup>  $\geq$  2, treatment will be re-initiated and continued until a vIGA-AD<sup>TM</sup> of 0 is achieved. This regimen of treatment and re-treatment will continue until the end of the study (i.e., subjects may receive study drug up until the Week 48 visit) (see Section 5.1.5.2 for additional details).

Study drug will be dispensed to subjects or their caregivers, applied during the clinic visits, and applied at home between clinic visits as instructed by site personnel. Subjects or their caregivers will be instructed to apply study drug QD to all affected areas, including newly appearing lesions and lesions/areas that improve during the study until a vIGA-AD<sup>TM</sup> of 0 is achieved. Once a vIGA-AD<sup>TM</sup> of 0 is achieved, the treatment period ends. If/when disease worsening occurs, and treatment is re-initiated at a vIGA-AD<sup>TM</sup> of  $\geq$  2, all lesions currently present and any new lesions that occur during the new treatment period should be treated.

Subjects or their caregivers will apply sufficient study drug to cover each lesion completely with a thin layer of study drug and will record the time of study drug application and daily itch score (PP-NRS) in a daily diary provided by the study site. Subjects are allowed, but not required, to treat scalp lesions with study drug; however, efficacy analyses will not include assessment of AD on the scalp. At the first clinic visit, if applicable, subjects and/or caregivers will be instructed to maintain the approximate dosing time for the daily application of study drug. At the phone contact at Week 2, subjects or caregivers should be reminded to complete their daily diary and bring it with them to the next clinic visit.


Clinical Study Protocol

Safety assessments will include AEs, clinical laboratory tests, physical examination, vital signs, and LTS. Efficacy assessments will include vIGA-AD<sup>TM</sup> score, %BSA affected, EASI, PP-NRS,

Refer to Section 6 for descriptions of study procedures and assessments and Section 7 and Table 1 for timing of procedures and assessments.

# 3.2 Treatment Groups and Duration

Subjects entering with a vIGA-AD<sup>TM</sup>  $\geq$  1 will receive treatment with tapinarof cream, 1% until they achieve a vIGA-AD<sup>TM</sup> score of 0, at which time treatment will be discontinued and subjects monitored for remittive effect. If/when disease worsening occurs, as evidenced by a vIGA-AD<sup>TM</sup>  $\geq$  2, treatment will then be re-initiated and continued until a vIGA-AD<sup>TM</sup> of 0 is achieved. Subjects entering with a vIGA-AD<sup>TM</sup> of 0 will have treatment discontinued beginning at the Baseline visit and will be monitored for remittive effect. If/when disease worsening occurs, as evidenced by a vIGA-AD<sup>TM</sup>  $\geq$  2, treatment will then be re-initiated and continued until a vIGA-AD<sup>TM</sup> of 0 is achieved. (Section 5.1.5.2 for additional details).

A subject will be considered to have completed the study when he/she completes all required procedures/visits for the 48-week treatment period and the Week 49 (Follow-Up) visit. The end of the study is defined as when the last active subject has completed the Follow-up Visit.

### 4 Study Population

# 4.1 Type and Number of Subjects

Up to 961 pediatric and adult subjects with AD will be enrolled in the study at up to approximately 135 study sites in the US and Canada.

Protocol violations from inclusion and exclusion criteria are prohibited because ineligible study subjects can potentially jeopardize the scientific integrity of the study, regulatory acceptability, or subject safety. Therefore, adherence to the criteria as specified in the protocol is essential.

#### 4.2 Inclusion Criteria

Each subject must meet all of the following criteria to be eligible to participate in the study:

# For Rollover Subjects Only:

- 1. Met the criteria as a Study Completer in one of three parent studies (Phase 3 pivotal safety and efficacy study DMVT-505-3101, Phase 3 pivotal safety and efficacy study DMVT-505-3102, or Phase 2 maximal use PK study DMVT-505-2104) and was still receiving study drug at the last visit of one of these studies.
  - NOTE: To meet the criteria as a Study Completer in one of the three parent studies, a subject must have completed  $\geq 80\%$  of the intended doses in that study.
- 2. Female subjects of childbearing potential must have a negative urine pregnancy test at Baseline (Day 1).

# For Direct-Enrolling Subjects Only:

- 3. Male and female subjects ages 2 years to < 18 years at the time of consent with clinical diagnosis of AD by Hanifin and Rajka criteria [Hanifin, 1980] (see Appendix 1).
- 4. Subjects with a vIGA-AD™ score of ≥ 3 and AD covering ≥ 40% of the BSA at Screening and Baseline (pre-randomization), or subjects with a vIGA-AD™ score of 2 at Screening and Baseline (pre-randomization) regardless of BSA. Scalp should be excluded from the BSA calculation to determine eligibility during Screening and at Baseline, and for all efficacy assessments. Subjects must have screened for the DMVT-505-3101 or DMVT-505-3102 study and failed to meet BSA and/or vIGA-AD™ eligibility criteria.
  - NOTE: Subjects with disease only on palms and soles are not eligible.
- 5. AD present for at least 6 months for ages 6 years old and above or 3 months for ages 2 to 5 years old, confirmed by prior medical documentation and/or according to the subject/caregiver report.
- 6. Female subjects of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test at Baseline (Day 1).

### For All Subjects (Rollover Subjects and Direct-Enrolling Subjects):

7. Female subjects of childbearing potential who are engaging in sexual activity that could lead to pregnancy should use one of the following acceptable birth control methods while on study and for 4 weeks after the last exposure to study drug.

• Acceptable contraception methods include intrauterine device, hormonal contraceptives, barrier method (e.g., condom or diaphragm), or surgical sterilization of male partner (vasectomy)


Clinical Study Protocol

- Subjects who claim abstinence as their method of contraception are allowed provided they agree to use a barrier method (e.g., condom or diaphragm) should they become sexually active from Baseline to 4 weeks after the last dose of study drug
  - Non-child-bearing potential is defined as:
- premenarchal
- pre-menopausal females with a documented bilateral tubal ligation, bilateral oophorectomy, hysterectomy, or hysteroscopic sterilization
- postmenopausal female with a cessation of menses for at least 12 months without an alternative medical cause; a blood sample with follicle stimulating hormone > 40 mIU/mL is confirmatory in questionable cases
- 8. Subject, subject's parent(s), or legal representative must be capable of giving written informed consent/assent, which includes compliance with the requirements and restrictions listed in the consent/assent form; written informed consent must be obtained prior to any study related procedures.

### 4.3 Exclusion Criteria

A subject who meets any of the following criteria will be excluded and considered ineligible for participation in the study:

# For Rollover Subjects Only:

- 1. Subjects who were not receiving study drug at the time of the last visit in the parent study (DMVT-505-3101, DMVT-505-3102, or DMVT-505-2104)
- 2. Used a prohibited concomitant product or procedure to treat AD during the parent study.
- 3. Had an SAE that was related to treatment or experienced an AE that led to permanent discontinuation of treatment in the parent study.
- 4. Pregnant females as determined by positive urine human chorionic gonadotropin test at Baseline.

# For Direct-Enrolling Subjects Only:

### 5. Concurrent conditions:

- a. Immunocompromised (e.g., lymphoma, acquired immunodeficiency syndrome) or medical history of positive human immunodeficiency virus antibody at Screening.
- b. Chronic or acute systemic infection requiring treatment with antiparasitics or antiprotozoals, within 4 weeks prior to the Baseline visit.
- c. Chronic or acute systemic bacterial infection requiring treatment with systemic antibiotics within one week prior to the Baseline visit.
- d. Chronic or acute superficial fungal infection requiring treatment with systemic antifungals within one week prior to the Baseline visit.
- e. Acute active bacterial, fungal, or viral (herpes simplex, herpes zoster, chicken pox) skin infection within 1 week prior to the Baseline visit; the condition should be completely resolved one week prior to Baseline Visit.

f. Significant dermatologic or inflammatory condition other than AD that, in the Investigator's opinion, would make it difficult to interpret data or assessments during the study. For example, subjects with an active skin condition such as Kaposi's varicelliform eruption, scabies, molluscum contagiosum, impetigo, psoriasis, severe acne, connective tissue disorder, or Netherton's syndrome, or any other concurrent active disease.

- g. Concurrent skin lesions in the treatment area or pruritus due to conditions other than AD that, in the opinion of the Investigator, would either interfere with study evaluations or affect the safety of the subject.
- 6. Screening alanine aminotransferase (ALT) or aspartate aminotransferase (AST)  $\geq$  2.0 x the upper limit of normal (ULN).
- 7. Screening total bilirubin > 1.5x ULN; total bilirubin > 1.5x ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%.
- 8. Current or chronic history of liver disease, known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones), presence of hepatitis B surface antigen (HBsAg), or positive hepatitis C antibody test result, or presence of anti-hepatitis B core antigen (anti-HBc). Subjects having a negative HBsAg and a positive anti-HBc may enroll if they have a positive anti-hepatitis B surface antigen demonstrating natural immunity. Subjects with a history of hepatitis C virus infection who were medically cured and have an undetectable viral load are eligible to enroll. Subjects with a history of stable non-alcoholic fatty liver disease without evidence of active inflammation (elevated ALT/AST ≥ 2.0x ULN) or cirrhosis are eligible to enroll.
- 9. Current or a history of cancer within 5 years except for adequately treated skin basal cell carcinoma, cutaneous squamous cell carcinoma or carcinoma in situ of the cervix (surgical excision or electrodessication and curettage).
- 10. Pregnant females as determined by positive serum (Screening) or urine (Baseline) human chorionic gonadotropin test.
- 11. Lactating females.
- 12. Previous known participation in a clinical study with tapinar of (previously known as GSK2894512 and WBI-1001).
- 13. Use of any prohibited medication or procedure within the indicated period before the Baseline visit.

NOTE: Prohibited concomitant medications, therapy, etc. during the defined period are as listed in the bullets below. If a subject requires any of these medications throughout the study period, he/she may be excluded from or discontinued from the study, at the discretion of the Investigator and Medical Monitor.

- a. From 4 months prior to Baseline:
  - o DUPIXENT® (dupilumab) injection.
  - Any monoclonal antibody product that becomes approved for AD during the course of the trial.

b. From 28 days prior to Baseline:

Oral, injectable, and suppository preparations of corticosteroids. Eye drops and nasal preparations are allowed. Inhaled preparations are allowed when used for a stable condition and stable dose for  $\geq 28$  days before Screening and are continued at the same dose throughout the study.


Clinical Study Protocol

- Oral preparations and injections of immunosuppressants (cyclosporine, methotrexate, azathioprine, tacrolimus, Janus kinase [JAK] inhibitors, etc.).
- Excessive sun exposure, tanning booth, other ultraviolet light source and phototherapy including psoralen and ultraviolet A therapy or is unwilling to minimize natural and artificial sunlight exposure.
- Treatment with antivirals with the exception of short-term treatment for acute upper respiratory viral infections (i.e., influenza) or viral suppressive therapy for a history of recurrent herpes labialis or genital herpes.

### c. From 14 days prior to Baseline:

- o EUCRISA® (crisaborole) and any other PDE4 inhibitor.
- o Tacrolimus ointment and pimecrolimus cream.
- Topical JAK inhibitors.
- Topical corticosteroids that are classified as medium or high potency (e.g., fluocinonide, triamcinolone acetonide) or super-high potency (e.g., clobetasol propionate). Eye drops and nasal preparations are allowed.
- Over the counter or herbal medicines for AD (topical and oral preparations). If subjects are using emollients, they may continue to use the same emollient on nonlesional skin during the study. Emollients containing salicylic acid are prohibited during the study.

### d. From 7 days prior to Baseline:

- Topical corticosteroids that are classified as low potency (e.g., desonide, hydrocortisone).
- o Oral, injectable, or intravenous antibiotics or antifungal medications.
- o Topical doxepin, topical gentamicin, or topical neomycin sulfate.
  - NOTE: Oral doxepin is allowed for treatment of depression if subject has been on a stable dose (4 weeks) at Screening
- o Topical products containing urea, except for the treatment of follicular events.
- Antihistamines/antiallergics (oral, topical and injections): diphenhydramine, chlorpheniramine maleate, hydroxyzine.

NOTE: For direct-enrolling subjects, the following antihistamines are allowed from Screening throughout the treatment period: loratedine, fexofenadine hydrochloride, cetirizine hydrochloride. Subjects are allowed to switch from non-allowed antihistamines to allowed antihistamines during Screening but must be on a stable dose for 7 days prior to Baseline.

e. The subject has received an investigational product within the following time period prior to the first dosing day in the current study: Minimum of 30 days or 5 half-lives of the investigational product (whichever is longer).

# For All Subjects (Rollover Subjects and Direct-Enrolling Subjects):

- 14. A history of or ongoing serious illness or medical, physical, or psychiatric condition(s) that, in the Investigator's opinion, may interfere with the subject's participation in the study, interpretation of results, safety of the subject or ability to understand and give informed consent.
- 15. Known hypersensitivity to tapinar of or excipients.

# 4.4 Lifestyle Restrictions

Subjects must avoid ultraviolet light, phototherapy, and excessive sun exposure throughout the study. When prolonged exposure cannot be avoided, use of sunscreen products (except on AD lesions) and protective apparel are recommended.

### 4.5 Withdrawal Criteria

A subject may voluntarily discontinue treatment and/or withdraw from participation in this study at any time at his/her own request or may be discontinued from study treatment at any time at the discretion of the Investigator for safety, behavioral, compliance, or administrative reasons. Subjects withdrawn from the study will not be replaced.

### 4.5.1 Reasons for Withdrawal from the Study

Study drug will be discontinued and the subject withdrawn from the study for any of the following reasons:

- Subject has an AE that is considered to be related to study drug or procedures AND is severe enough to warrant treatment discontinuation, as determined by the Investigator (Section 8.1).
- Pregnancy
- Any Grade 3 or 4 AE, based on Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) criteria, considered causally related to study drug (Section 8.2.2)

Study drug may be discontinued and the subject withdrawn from the study for any of the following reasons:

- Subject requires concurrent prohibited medication during the study (Section 5.6.2). Nonmedicated emollients that do not contain salicylic acid may be used on nonlesional skin but the subject (or caregiver) should wait at least 30 minutes after applying study drug before applying nonmedicated emollients; emollients should not be applied to lesional skin during treatment. The same emollient should be used throughout the subject's participation in the study.
  - NOTE: If, in the opinion of the Investigator and the study Medical Monitor, such medication will not interfere with the conduct or interpretation of the study or compromise the safety of the subject, then the subject may continue to receive study drug.
- Subject noncompliance
- Investigator noncompliance
- Discontinuation of the study at the request of the Sponsor, regulatory agency, or an Institutional Review Board (IRB)/Independent Ethics Committee (IEC).

If a subject meets a withdrawal criterion during treatment, an Early Termination visit will be required (Section 7.7).

### 4.5.2 Withdrawal Procedures

The primary reason for the discontinuation of study drug and/or withdrawal from study must be recorded in the source document and on the case report form (CRF). If a subject is prematurely discontinued from study drug, the Investigator must make every effort to perform an Early Termination Visit (Section 7.7) and document the primary reason for withdrawal.

### 4.6 Lost to Follow-Up

A subject is considered lost to follow-up if he/she repeatedly fails to return to the study site for scheduled visits and is unable to be contacted by the study site. The following actions must be taken if a subject fails to return to the clinic for a required study visit:

- The site must attempt to contact the subject or caregiver and reschedule the missed visit as soon as possible, counsel the subject and/or caregiver on the importance of maintaining the assigned visit schedule, and ascertain whether or not the subject wishes to and/or should continue in the study.
- Before a subject is deemed lost to follow-up, the Investigator or designee must make every effort to regain contact with the subject or caregiver (where possible, 3 telephone calls and, if necessary, a certified letter to the subject's last known mailing address or local equivalent methods). These contact attempts should be documented in the subject's medical record.
- Should the subject or caregiver continue to be unreachable, he/she will be considered to have withdrawn from the study with a primary reason of lost to follow-up. In this case, the discontinuation date will be listed as the date the certified letter was mailed to the subject.
# 5 Study Treatment

# 5.1 Study Drug

# 5.1.1 Description, Packaging, and Labeling

The description of the study drug, tapinar of cream, 1%, is presented in Table 2.

Table 2: Tapinar of Cream



All labels for tapinar of cream, 1% to be distributed in the participating countries will meet all applicable requirements of those countries.

# 5.1.2 Storage

All study drugs must be stored in a secure environmentally controlled and monitored (manual or automated) area in accordance with the labeled storage conditions, with access limited to the Investigator and authorized site staff. The study drug storage temperature range will be provided in the Study Reference Manual.

# 5.1.3 Handling and Disposal

Under normal conditions of handling and administration, study drug is not expected to pose significant safety risks to site staff. In the case of unintentional occupational exposure notify the monitor, Medical Monitor and/or the Sponsor study contact.

Arrangements will be made for used and unused drug supplies to be returned to the Sponsor or Sponsor designee, or for destruction on site following acceptable, documented procedures. Further guidance and information for final disposition of unused study drug will be provided.

# 5.1.4 Preparation

No special preparation of study drug is required.

# 5.1.5 Administration of Study Drug

# 5.1.5.1 Treatment Based on Validated Investigator Global Assessment of Atopic Dermatitis

Subjects entering with a vIGA-AD<sup>TM</sup>  $\geq$  1 (including all subjects enrolling directly into this study) will receive treatment QD with tapinarof cream, 1% until they achieve a vIGA-AD<sup>TM</sup> score of 0, at which time treatment will be discontinued and subjects monitored for maintenance of disease control (i.e. the extent of the remittive effect). If/when disease worsening occurs, as evidenced by a flare to vIGA-AD<sup>TM</sup>  $\geq$  2, treatment will be reinitiated and continued until a vIGA-AD<sup>TM</sup> of 0 is achieved. Subjects entering with a vIGA-AD<sup>TM</sup> of 0 will

have treatment discontinued beginning at the Baseline visit and will be monitored for maintenance of the remittive effect. If/when disease worsening occurs, as evidenced by a flare to vIGA-AD<sup>TM</sup>  $\geq$  2, treatment will be re-initiated and continued until a vIGA-AD<sup>TM</sup> of 0 is achieve. Once a vIGA-AD<sup>TM</sup> of 0 is achieved, the treatment period ends. If/when disease worsening occurs, and treatment is re-initiated at a vIGA-AD<sup>TM</sup> of  $\geq$  2, all lesions currently present and any new lesions that occur during the new treatment period should be treated. This treatment and re-treatment pattern of use will be continued until the end of the study (i.e., subjects may receive study treatment up until the Week 48 visit).

Subjects who experience suspected disease worsening between scheduled study visits may contact the study site to arrange an unscheduled visit (Section 7.6). See Section 5.1.5.2 for further instructions. Upon confirmation of disease worsening, subjects will restart treatment with study drug.

# 5.1.5.2 Disease Worsening (Validated Investigator Global Assessment of Atopic Dermatitis ≥ 2 During the Study)

If disease worsening is suspected between scheduled study visits, an unscheduled visit may be performed. If disease worsening (i.e.,  $vIGA-AD^{TM} \ge 2$ ) is not confirmed, the subject will continue to be assessed at routine, scheduled visits (see Table 1).

For each confirmed episode of disease worsening (i.e., vIGA-AD<sup>TM</sup>  $\geq$  2) during the study (at either a scheduled or unscheduled visit), a treatment course of tapinarof cream, 1% QD will be initiated and will continue until the subject achieves a vIGA-AD<sup>TM</sup> of 0, as assessed at scheduled visits, approximately every 4 weeks beginning at Baseline.

# 5.1.5.3 Application of Study Drug

Study drug will be dispensed to subjects or their caregivers at the clinical site in appropriately labeled tubes.

Subjects or caregivers will take the tubes home and self-administer study drug (or have caregiver apply if necessary) to affected areas QD, except on clinic visit days when study drug is applied under supervision at the site.

Subjects will be instructed to apply study drug as follows:

- QD application to affected areas; subjects or their caregivers are advised to choose the application time they prefer and to apply the study drug at that approximate time each day of study participation. Subjects should avoid dosing around midnight to avoid potentially dosing twice in one calendar day.
- If a subject misses a daily dose, it will be recorded as a protocol deviation. The subject should continue dosing the next day and should not apply more than once daily to make up for the missed dose on the previous day. If a dose is missed, the missed dose and the reason for the missed dose should be recorded in the daily diary as such. Itch rating can still be recorded in the diary even if a daily dose was missed.
- Study drug should be applied to dry, clean skin.
- Study drug may be applied to skin around the eye but avoid direct contact with the eye study drug is not for ophthalmic use.
- Wash hands after application, unless treating lesions on the hands.

• Study drug should be applied to all lesions, including newly appearing lesions and lesions/areas that improve during the study until a vIGA-AD<sup>TM</sup> of 0 is achieved. Once a vIGA-AD<sup>TM</sup> of 0 is achieved, the treatment period ends. If/when disease worsening occurs, and treatment is reinitiated at a vIGA-AD<sup>TM</sup> of ≥ 2, all lesions currently present and any new lesions that occur during the new treatment period should be treated. A body diagram identifying locations of lesions may be provided to the subject and/or caregiver.


Clinical Study Protocol

- Subjects are allowed, but not required, to treat scalp lesions with study drug; however, efficacy analyses will not include assessment of AD in this area.
- If there is residual cream visible on the disease-affected lesional skin, then the subject or caregiver should be instructed to continue to lightly rub the cream into the skin until it is no longer visible.
- If study drug is applied to the subject by another person, that person should thoroughly wash his/her hands after application.
- When dosing at home subjects or caregiver should record the time of study drug application in the daily diary. Itch rating should also be recorded in the diary.
- On clinic visit days, study drug should be applied in the clinic under the supervision of site personnel and after safety and efficacy assessments have been completed

NOTE: The time of the dose and assessments on clinic visit days will depend on the time of the clinic visit. Therefore, the timing of the clinic visit may differ from the subject's chosen dosing time. The intention is to allow flexibility to accommodate subjects' schedules.

• Nonmedicated emollients that do not contain salicylic acid may be used on nonlesional skin but the subject (or caregiver) should wait at least 30 minutes after applying study drug before applying nonmedicated emollients; emollients should not be applied to lesional skin during treatment. The same emollient should be used throughout the subject's participation in the study.



#### 5.2 Randomization/Treatment Assignment

All subjects will receive treatment with tapinar of cream, 1% as needed per protocol.

# 5.3 Blinding

This study is an open-label study; blinding is not applicable.

# 5.4 Compliance with Study Drug Administration

At Baseline, study staff will provide the subject or caregiver with detailed instructions concerning protocol requirements and use of study drug. Additionally, subjects or caregivers will be asked to complete a daily diary with the time of each application of study drug, except on study visit days. At each post-Baseline study visit, study staff will review use of study drug, as applicable, with the subject or caregiver. Subject compliance will be assessed via study diary completion.

When subjects are dosed at the site, they and/or their caregiver will apply the study drug under supervision of the study staff. The date and time of each dose administered in the clinic will be recorded in the source documents. The study drug and study subject identification should be confirmed at the time of dosing by a member of the study site staff other than the person dispensing the study drug.

At the time of dispensing study drug to each subject, site personnel will weigh the tubes to be dispensed with the cap on and will record the weight of all tubes dispensed at each visit in the drug accountability logs. Subjects and/or caregivers will be instructed to bring all used and unused tubes with them to each study visit. Site personnel will weigh the returned tubes (used and unused) with the cap on and record the weight in the drug accountability logs. If a tube has been lost, discarded, or forgotten by the subject, then the site personnel will make a notation of this on the drug accountability logs. Forgotten tubes should be returned by the subject at the next study visit. Tubes of study medication dispensed at the most recent prior visit which remain unopened (the foil cap on the tube remains fully intact/undisturbed) may be re-dispensed to study subjects at the current visit. Unopened tubes may only be re-dispensed once. Opened, partially used tubes or tubes with foil overlay removed are not to be re-dispensed to study subjects. If there is any question as to re-dispensation, sites should issue new tubes of study medication to the subject(s).

# 5.5 Treatment after the End of the Study

Subjects will not receive any additional treatment with the study drug from the Sponsor after completion of the study because the indication being studied is not life threatening or seriously debilitating and other treatment options are available.

The Investigator is responsible for ensuring that consideration has been given to the post study care of the subject's medical condition, whether or not the Sponsor is providing specific post-study drug.

# 5.6 Prior and Concomitant Therapy

For rollover subjects, any medication (including over the counter or prescription medication, vitamins and/or herbal supplements) administered to the subject at the time of enrollment and during the study must be recorded on the CRF along with the reason for use. For direct-enrolling subjects, any medication (including over the counter or prescription medication, vitamins and/or herbal supplements) administered to the subject up to 30 days before the Screening visit, at the time of enrollment, and during the study must be recorded in the CRF along with the reason for use. The information to be recorded must also include name of the medication (generic name, as a general rule), dose, frequency, administration routes, and dates of the first and last dose, as applicable.

The Medical Monitor should be contacted if there are any questions regarding concomitant or prior therapy.

# 5.6.1 Permitted Medications and Nondrug Therapies

Concomitant medications for medical treatment of other conditions are allowed under the condition that the dosage and administration of these treatments is not planned to change from the Baseline visit to the completion of the treatment phase (Week 48) and that the medication is not a prohibited medication as described in the Exclusion Criteria (Section 5.6.2).

In the event of skin infection, topical antibacterial agents with the exception of gentamicin and neomycin sulfate can be applied to the infected area; however, study drug must not be applied to the area until the skin infection is healed.

Nonmedicated emollients that do not contain salicylic acid may be used on nonlesional skin but the subject (or caregiver) should wait at least 30 minutes after applying study drug before applying nonmedicated emollients; emollients should not be applied to lesional skin during treatment. The same emollient should be used throughout the subject's participation in the study.

Any emollient used during the study must be recorded as a concomitant medication.

# 5.6.2 Prohibited Medications and Nondrug Therapies

Medications and nondrug therapies that are prohibited throughout the study duration are as follows:

- DUPIXENT® (dupilumab) injection, or any monoclonal antibody product that becomes approved for AD during the course of the trial
- Oral, injectable, and suppository preparations of corticosteroids. Eye drops and nasal preparations are allowed. Inhaled preparations are allowed when used for a stable condition and stable dose for > 28 days before Baseline and are continued at the same dose throughout the study.
- Oral preparations and injections of immunosuppressants (cyclosporine, methotrexate, azathioprine, tacrolimus, JAK inhibitors, etc.).
- Excessive sun exposure, tanning booth, other ultraviolet light source and phototherapy including psoralen and ultraviolet A therapy or is unwilling to minimize natural and artificial sunlight exposure.
- Treatment with antivirals with the exception of short-term treatment for acute upper respiratory viral infections (i.e., influenza) or viral suppressive therapy for a history of recurrent herpes labialis or genital herpes.
- EUCRISA® (crisaborole) and any other phosphodiesterase 4 inhibitor.
- Tacrolimus ointment and pimecrolimus cream.
- Topical JAK inhibitors.
- Topical corticosteroids that are classified as low potency (e.g., desonide, hydrocortisone), medium or high potency (e.g., fluocinonide, triamcinolone acetonide) or super-high potency (e.g., clobetasol propionate). Eye drops and nasal preparations are allowed.
- Over the counter or herbal medicines for AD (topical and oral preparations). If subjects are using emollients, they may continue to use the same emollient on nonlesional skin during the study. Emollients containing salicylic acid are prohibited during the study.
- Oral, injectable, or intravenous antibiotics or antifungal medications.

• Topical doxepin or topical antibiotics.

NOTE: Oral doxepin is allowed for treatment of depression if subject has been on a stable dose (4 weeks) at Screening

• Antihistamines/antiallergics (oral, topical and injections): diphenhydramine, chlorpheniramine maleate, hydroxyzine.

NOTE: The following antihistamines are allowed from Screening throughout the treatment period: loratadine, fexofenadine hydrochloride, cetirizine hydrochloride. Subjects are allowed to switch from non-allowed antihistamines to allowed antihistamines during Screening but must be on a stable dose for 7 days prior to Baseline.

Any investigational products or procedures.

A list of prohibited medications, emollients and nondrug therapies may be provided as a separate document. If a subject chooses to treat scalp with study drug, then medicated shampoos are prohibited for use. Emollients containing salicylic acid are prohibited.

## **6 Study Assessments and Procedures**

Study procedures and assessments are summarized in the Schedule of Assessments (Table 1) and in Section 7. Adherence to the study design requirements, including those specified in the Schedule of Assessments are essential and required for study conduct. Protocol waivers or exemptions are not allowed, except for immediate safety concerns.

For rollover subjects, age is determined as age at the time of consent in the parent study. For direct-enrolling subjects, age is determined as age at the time of consent in this study. In both cases, the determined age will remain the same throughout the duration of this study for the purposes of completing all study assessments.

# 6.1 Medical History, Demography, and Baseline Characteristics

# 6.1.1 Demographics

For rollover subjects, demographic information collected during the parent study will be used for this study, including age, sex, race, and ethnicity.

For direct-enrolling subjects, demographic information collected will include age, sex, race, ethnicity, and Fitzpatrick skin type. Information on Fitzpatrick skin type can be found in Appendix 2.

#### **6.1.2** Medical History

For rollover subjects, medical, medication, and family history collected during the parent study will be used for this study.

For direct-enrolling subjects, Medical history will be collected to ensure subjects are eligible for participation in the study per inclusion (Section 4.2) and exclusion (Section 4.3) criteria. Data collected for direct-enrolling subjects will include year of AD diagnosis, allergic conditions, cardiovascular (CV) medical history and risk factors (including height, weight, blood pressure, medical conditions, and family history of premature CV disease), and family history of liver disease. As part of the direct-enrolling subject's medical history, all systemic (oral and injectable) medications used by the subject for treatment of AD prior to 30 days before the Screening visit will be collected.

For all subjects (rollover subjects and direct-enrolling subjects), if a subject has previously tested positive for COVID-19 or has previously received a COVID-19 vaccine, it should be documented in the subject's medical history.

## 6.2 Safety Assessments

#### **6.2.1** Adverse Events

All AEs and SAEs will be collected from the time the subject signs the informed consent form (ICF) until the final visit/contact with the subject. AEs that began during the parent study and were ongoing at the end of that study will be reported as ongoing AEs. Additional safety information, including the definition of an AE and the methods for recording, evaluating, and assessing causality of AEs and the procedures for completing and transmitting SAE reports are provided in Section 8.

# **6.2.2** Brief Physical Examination

A brief physical examination will include, at a minimum, assessments of the skin, lungs, cardiovascular system, and abdomen (liver and spleen). Assess for changes in onset of menses (female participants) or sexual activity (male or female participants). Determine if there is a need for contraception or barrier use. Investigators should pay special attention to clinical signs related to previous serious illness.

For direct-enrolling subjects, height and weight will be measured at Screening only.

# 6.2.3 Vital Signs

Vital signs will be measured before blood collection for clinical laboratory assessments and will include measurements of systolic and diastolic blood pressure, pulse rate, and body temperature. Subjects should be in a seated position for at least 5 minutes before vital signs measurement.


Clinical Study Protocol

# **6.2.4** Clinical Safety Laboratory Assessments

All protocol-required laboratory assessments must be conducted in accordance with the Study Reference Manual or Laboratory Manual and the protocol Schedule of Assessments (Table 1). Laboratory requisition forms must be completed, and samples must be clearly labeled with the subject number, protocol number, site number, and visit date. Details for the preparation and shipment of samples will be provided by the laboratory and are detailed in the Study Reference Manual or the Laboratory Manual. Reference ranges for all safety parameters will be provided to the site by the laboratory responsible for the assessments.

A list of clinical laboratory tests and parameters is provided in Table 3.

All laboratory tests with values that are considered clinically significantly abnormal during participation in the study should be repeated until the values return to normal or Baseline. If such values do not return to normal within a period judged reasonable by the Investigator, the etiology should be identified, if possible, and the Sponsor and Medical Monitor notified.

#### **Table 3:** Laboratory Tests

# Diagnostic Tests

- All subjects
  - Urine pregnancy tests (WOCBP only)<sup>a</sup>
- <u>Direct-Enrolling Subjects Only</u>
  - Serum pregnancy test at Screening (WOCBP only)
  - HBsAs
  - Hepatitis C antibody
  - Anti-HBc
  - Anti-HBs<sup>b</sup>
  - At the Investigator's discretion, subjects may be screened for alcohol and illicit drug use.

| Serum Chemistry | | |
|---|---|---|
| • BUN | Total carbon dioxide | Uric acid |
| Creatinine | Calcium | • Total bilirubin (+fractionated if |
| Glucose (fasting not required) | • AST | required) |
| Sodium | • ALT | Total protein |
| Potassium | Alkaline phosphatase | Albumin |
| Chloride | | |
| Hematology | | |
| Platelet count | RBC Indices: | • WBC Differential: |
| RBC count | • MCV | <ul> <li>Neutrophils</li> </ul> |
| WBC count (absolute) | • MCH | <ul> <li>Lymphocytes</li> </ul> |
| Reticulocyte count | • MCHC | <ul> <li>Monocytes</li> </ul> |
| Hemoglobin | Reticulocyte percentage | <ul> <li>Eosinophils</li> </ul> |
| Hematocrit | | <ul> <li>Basophils</li> </ul> |

| Definition Sciences, inc. | |
|---|---|
| Urinalysis | |
| Specific gravity | <u>Dipstick</u> : pH, Glucose, Protein, Blood |
| Microscopic examination (if blood or protein is abnormal) | Ketones |

- a. Pregnancy tests should be administered based on CBP, which may change after the start of the study (e.g. a premenarchal female subject experiences menarche or a female subject ceases to meet the criteria of CBP)
- b. Reflex test: a negative HBsAg and a positive anti-HBc may enroll if there is a positive anti-HBs demonstrating natural immunity ALT = alanine aminotransferase; Anti-HBc = anti-hepatitis B core antigen; Anti-HBs = anti-hepatitis B surface antigen;
- AST = aspartate aminotransferase; BUN = blood urea nitrogen; HBsAg = hepatitis B surface antigen; MCH = mean corpuscular hemoglobin; MCHC = mean corpuscular hemoglobin concentration; MCV = mean corpuscular volume; RBC = red blood cell(s); WBC = white blood cell(s); WOCBP = women of child-bearing potential



### 6.3 Efficacy Assessments

To minimize inter observer variability, Investigators and/or evaluators/raters will be trained on each of the required assessments during an Investigator meeting, site initiation visit, and/or utilizing online assessments before enrolling subjects at their study site. Only trained evaluators/raters are permitted to perform the efficacy assessments. To the fullest extent possible, the same Investigator (or designated evaluator/rater) will perform all efficacy assessments for an individual subject throughout the study. If it is not possible for the same evaluator/rater to continue performing assessments, it is recommended that the primary and subsequent evaluator/rater both examine and discuss their respective scoring during at least 1 visit.

# 6.3.1 Assessments Completed by Investigator

## 6.3.1.1 Validated Investigator Global Assessment of Atopic Dermatitis

The vIGA-AD<sup>TM</sup> of disease severity will be assessed at every clinic visit. The vIGA-AD<sup>TM</sup> is a global assessment of the current state of the disease. It is a 5-point morphological assessment of overall disease severity (scalp excluded) and will be determined according to the categories described in Table 4 and Appendix 5. Eli Lilly and Company developed the vIGA-AD<sup>TM</sup> scale for use in clinical trials.

| Table 4: | Validated Investigator | Global Assessment | Scale for Ato | pic Dermatitis |
|---|---|---|---|---|

| Score | Category | Definition |
|---|---|---|
| 0 | Clear | No inflammatory signs of atopic dermatitis (no erythema, no induration/papulation, no lichenification, no oozing/crusting). Post-inflammatory hyperpigmentation and/or hypopigmentation may be present. |
| 1 | Almost clear | Barely perceptible erythema, barely perceptible induration/papulation, and/or minimal lichenification. No oozing or crusting. |
| 2 | Mild | Slight but definite erythema (pink), slight but definite induration/papulation, and/or slight but definite lichenification. No oozing or crusting |
| 3 | Moderate | Clearly perceptible erythema (dull red), clearly perceptible induration/papulation, and/or clearly perceptible lichenification. Oozing and crusting may be present. |
| 4 | Severe | Marked erythema (deep or bright red), marked induration/papulation, and/or marked lichenification. Disease is widespread in extent. Oozing or crusting may be present. |

# 6.3.1.2 Body Surface Area Affected

The assessment of the %BSA affected is an estimate of the percentage of total involved skin with AD. For the purpose of clinical estimation, the total palmar surface of the subject's palm and digits may be assumed to be approximately equivalent to 1% BSA. The %BSA affected by AD will be evaluated from 0% to approximately 100% (scalp excluded). Details on calculation of approximate %BSA involvement in each subject are provided in Appendix 6. Percentage BSA is a static assessment made without reference to previous scores.

# 6.3.1.3 Eczema Area and Severity Index

The EASI will be assessed at every clinic visit. It quantifies the severity of a subject's AD based on both lesion severity and the %BSA affected [Hanifin, 2001]. The subject's scalp is excluded from this assessment. The EASI is a composite score ranging from 0 to 72 that takes into account the degree of erythema, edema/papulation, excoriation, and lichenification (each scored from 0 to 3 separately) for each of four body

regions, with adjustment for the %BSA involved for each body region relative to the whole body. A detailed procedure of EASI score calculation is provided in Appendix 6. The EASI score will be calculated in the CRF based on the subject's age, the rating scores for each region, and the number of handprints involved for each region.

# 6.3.2 Assessments Completed by Subject or Caregiver

A summary table of assessments completed by subject or caregiver, broken down by age group, is provided in Appendix 7.



# 6.3.2.3 Peak Pruritus-Numeric Rating Scale

The PP-NRS is a scale used to quickly assess itch/pruritus severity over a 24-hour period. The subject or caregiver will utilize the scale to assess peak pruritus QD and record the results in their daily diaries. The itch

rating can be done before or after study drug administration since it should reflect the past 24 hours. On clinic visit days, the PP-NRS will be assessed in the clinic. PP-NRS should be completed every day, even if subjects are not actively applying study drug. For subjects ages 2 to < 12 years, the PP-NRS will be completed by the caregiver. For subjects ages  $\geq$  12 years, the PP-NRS will be completed by the subject.

An example of the PP-NRS is provided in Appendix 13.





# 6.3.3 Optional Clinical Photography

Clinical photography may be performed in a subgroup of subjects at selected study sites. Informed consent/assent and photographic release will be required. The photographs may not be referred to by the Investigator at any subsequent study visit for the purposes of grading.

Photographs will be taken of a representative area of the subject's disease area at the time points specified in the Schedule of Assessments (Table 1). Photographs of the selected skin area will be taken in a standardized fashion (i.e., same camera, angle, background, distance).

# 6.4 Treatment of Study Drug Overdose

For this study, accidental or intentional oral ingestion of drug product will be considered an overdose. Ingestion of a 30-gram tube of tapinar fcream, 1% would result in an oral dose of 300 mg.

The Sponsor does not recommend specific treatment for an overdose; however, in the event of an overdose, the Investigator (or treating physician) should do the following:

- Contact Medical Monitor to discuss the event
- Closely monitor the subject for AEs/SAEs and laboratory abnormalities
- Provide general symptomatic treatment as necessary
- Document the quantity of the excess dose as well as the duration of the overdosing.

Decisions regarding dose interruptions or modifications following an overdose will be made by the Investigator in consultation with the Medical Monitor based on the clinical evaluation of the subject.

#### **6.5** Virtual Assessments

In the event that a subject cannot attend their regularly scheduled study visits in person <u>due to a COVID-19-like situation necessitating a limit on in-person contact</u>, the Investigator may perform safety and efficacy assessments by phone or video. Source documentation should note if the visit was performed by phone or by video. The Investigator may use the technology platform that is currently available to them. Suggested platforms include Apple FaceTime, Zoom for Healthcare, Facebook Messenger video chat, Microsoft Teams, Google Hangouts video, and Skype. Additional details of the visit should be included in source documentation, as detailed in the Study Reference Manual.

If the subject can only be contacted by phone, the following should be assessed or performed:

- AEs
- Concomitant Medications
- Reminder to complete diary
- Instruction not to discard empty tubes of study drug

If the subject has video capabilities, the following items should be assessed or performed:

- AEs
- Concomitant Medications
- vIGA-AD<sup>TM</sup> assessment (excluding subject's scalp)
- %BSA assessment (excluding subject's scalp)
- EASI (excluding subject's scalp)
- •
- Application of study drug by the subject or caregiver, if applicable
   Completion of the RP NPS (the subject or caregiver [or applicable] care
- Completion of the PP-NRS (the subject or caregiver [as applicable] can verbally indicate the answer which the study coordinator will document in the source document).


Clinical Study Protocol

- Reminder to complete diary
- Instruction not to discard empty tubes of study drug

The reason that assessments cannot be completed during a virtual assessment (i.e., labs, vital signs, physical exams, etc.) must be noted (e.g., COVID-19) and the missed assessments will be recorded as protocol deviations.

## 7 Timing of Procedures and Assessments

This section lists the procedures and assessment to be performed at scheduled time points during the study as outlined in the Schedule of Assessments (Table 1). Information on study procedures and assessments is provided in Section 6.

- Any change in timing or any addition of a time point(s) for any planned study assessment must be documented in a "Note to File," which is approved by the relevant Sponsor study team member and then archived in the study Sponsor and site study files; this will NOT constitute a protocol amendment.
- The IRB/IEC will be informed of any safety issues that require alteration of the safety monitoring or amendment of the ICF.

# 7.1 Visit 0; Screening Period for Direct-Enrolling Subjects (Day -30 to Day -1)

After the subject has signed the consent/assent form, potential study subjects will undergo Screening procedures and assessments to confirm eligibility to participate in the study. Screening assessments will include the following:

- Demography recording
- Fitzpatrick skin type
- Medical history recording
- Brief physical examination (including height and weight, body mass index will be calculated in the CRF)
- Vital signs measurements
- Serum pregnancy test (women of child-bearing potential [WOCBP])
- Blood sample collection for clinical laboratory tests (serum chemistry, hematology, diagnostic tests)
- Urinalysis
- vIGA-AD<sup>TM</sup> score (excluding subject's scalp)
- %BSA affected calculation (excluding subject's scalp)
- EASI (excluding subject's scalp)
- AE recording (from the time the ICF is signed)
- Concomitant medication recording (including all medications administered up to 30 days prior to screening, and all systemic [oral and injectable] medications used by the subject for the treatment of AD prior to 30 days before Screening)

## 7.2 Visit 1; Baseline (Day 1)

# 7.2.1 Baseline Visit for Subjects Rolling Over from DMVT-505-3101 and DMVT-505-3102

On Day 1, subjects from the parent studies DMVT-505-3101 or DMVT-505-3102 who were considered eligible for this study will sign the ICF and be reassessed to confirm eligibility to participate in this study. All subjects who continue to meet study eligibility criteria will be enrolled. Subjects entering with a vIGA-AD<sup>TM</sup>  $\geq$  1 will receive treatment with tapinar of cream, 1% until they achieve a vIGA-AD<sup>TM</sup> score of 0, at which time treatment will be discontinued and subjects monitored for maintenance of the remittive effect. If/when

disease worsening occurs, as evidenced by a vIGA-AD<sup>TM</sup>  $\geq$  2, treatment will then be re-initiated and continued until a vIGA-AD<sup>TM</sup> of 0 is observed. Subjects entering with a vIGA-AD<sup>TM</sup> of 0 will have treatment discontinued beginning at the Baseline visit and will be monitored for maintenance of the remittive effect.

The following procedures and assessments will be performed at the Baseline visit:

- Demographics and Fitzpatrick skin type (carried over from parent study)
- Medical history (carried over from parent study)
- Brief physical exam (last assessment from parent study)
- Vital signs measurements (last assessment from parent study)
- Urine pregnancy test (WOCBP; last assessment from parent study)
- Blood sample collection for clinical laboratory tests (serum chemistry and hematology; last assessment from parent study)
- Urinalysis (last assessment from parent study)
- vIGA-AD<sup>TM</sup> score (excluding subject's scalp; last assessment from parent study)
- %BSA affected calculation (excluding subject's scalp; last assessment from parent study)
- EASI (excluding subject's scalp; last assessment from parent study)
- PP-NRS (last assessment from parent study)
  Image: PP-NRS (last assessment from parent study)
- Photography of a representative area of the subject's disease area (at a subset of study sites only; last photograph from parent study)
- AE recording (ongoing from parent study at the time the ICF is signed in this study)
- Concomitant medication recording (ongoing from parent study at the time the ICF is signed in this study)
- Dispense diary (subjects or their caregivers will be instructed in how and when to complete diary)
- Dispense study drug, if applicable
- Instruction on how to apply study drug, if applicable
- Study drug application under supervision, if applicable

# 7.2.2 Baseline Visit for Subjects Rolling Over from DMVT-505-2104

On Day 1, subjects from the parent studies DMVT-505-2104 who were considered eligible for this study will sign the ICF and be reassessed to confirm eligibility to participate in this study. All subjects who continue to meet study eligibility criteria will be enrolled. Subjects entering with a vIGA-AD<sup>TM</sup>  $\geq$  1 will receive treatment with tapinarof cream, 1% until they achieve a vIGA-AD<sup>TM</sup> score of 0, at which time treatment will be discontinued and subjects monitored for maintenance of the remittive effect. If/when disease worsening

occurs, as evidenced by a vIGA-AD<sup>TM</sup>  $\geq$  2, treatment will then be re-initiated and continued until a vIGA-AD<sup>TM</sup> of 0 is observed. Subjects entering with a vIGA-AD<sup>TM</sup> of 0 will have treatment discontinued beginning at the Baseline visit and will be monitored for maintenance of the remittive effect.

The following procedures and assessments will be performed at the Baseline visit:

- Demographics and Fitzpatrick skin type (carried over from parent study)
- Medical history (carried over from parent study)
- Brief physical exam (last assessment from parent study)
- Vital signs measurements (last assessment from parent study)
- Urine pregnancy test (WOCBP; last assessment from parent study)
- Blood sample collection for clinical laboratory tests (serum chemistry and hematology; last assessment from parent study)
- Urinalysis (last assessment from parent study)
- vIGA-AD<sup>TM</sup> score (excluding subject's scalp; last assessment from parent study)
- %BSA affected calculation (excluding subject's scalp; last assessment from parent study)
- EASI (excluding subject's scalp; last assessment from parent study)



- AE recording (ongoing from parent study at the time the ICF is signed in this study)
- Concomitant medication recording (ongoing from parent study at the time the ICF is signed in this study)
- Dispense diary (subjects or their caregivers will be instructed in how and when to complete diary)
- Dispense study drug, if applicable
- Instruction on how to apply study drug, if applicable
- Study drug application under supervision, if applicable

## 7.2.3 Baseline Visit for Subjects Enrolling Directly into DMVT-505-3103

On Day 1, subjects will be reassessed to confirm continued eligibility to participate in the study. All subjects who continue to meet study eligibility criteria will be randomized to treatment.

The following additional procedures and assessments will be performed at the Baseline Visit:

- Changes to medical history will be recorded
- Brief physical examination
- Vital signs measurement
- Urine pregnancy test (WOCBP)

• Blood sample collection for clinical laboratory tests (serum chemistry and hematology)

NOTE: Blood sample collection for clinical laboratory tests is not required at the Baseline Visit if it has been  $\leq$ 14 days since samples were collected at Screening and the results of those clinical laboratory tests were within the normal range.

• Urinalysis

NOTE: Urine sample collection for urinalysis is not required at the Baseline Visit if it has been ≤14 days since samples were collected at Screening and the results of those analyses were within the normal range.

- vIGA-AD<sup>TM</sup> score (excluding subject's scalp)
- %BSA affected calculation (excluding subject's scalp)
- EASI (excluding subject's scalp)



- Photography of a representative area of the subject's disease area (at a subset of study sites only)
- AE recording
- Concomitant medication recording
- Dispense diary (subjects or their caregivers will be instructed on how and when to complete diary)
- Dispense study drug
- Instruction on how to apply study drug
- Study drug application under supervision

#### 7.3 Visits 2 to 13; Treatment Period

Subjects will return to the study site at least every 4 weeks ( $\pm 3$  days) during the 48-week monitoring period. The following assessments will be performed:

- Brief physical exam; Weeks 12, 24, 36 and 48 only
- Vital signs measurements
- Urine pregnancy test (WOCBP)
- Blood sample collection for clinical laboratory tests (serum chemistry and hematology); Weeks 12, 24, 36 and 48 only
- Urinalysis; Week 48 only
- vIGA-AD<sup>TM</sup> score (excluding subject's scalp)
- %BSA affected calculation (excluding subject's scalp)
- EASI (excluding subject's scalp)

PP-NRS (by subject or caregiver)


- Photography of a representative area of the subject's disease area (at a subset of study sites only); Weeks 12, 24, 36 and 48 only
- AE recording
- Concomitant medication recording
- Collect and review subject diaries for treatment compliance
- Dispense diary
- Collect and dispense study drug, if applicable
- Review instructions on how to apply study drug, if applicable
- Study drug application under supervision, if applicable

# 7.4 Phone Contact at Week 2 (Day $15 \pm 3$ Days)

Subjects or their caregivers will be contacted by phone at Week 2 to review study drug application instructions, if applicable, and to record AEs and concomitant medication use. Subjects or their caregivers should be reminded to complete their daily diary and bring it with them to the next clinic visit.

# 7.5 Follow-Up Visit 14; Week 49 (Day $344 \pm 3$ Days)

Subjects will return to the study site 1 week ( $\pm 3$  days) after last treatment to complete follow-up assessments as follows:

- Brief physical examination
- Vital signs measurement
- Blood sample collection for clinical laboratory tests (serum chemistry and hematology)
- Urinalysis
- vIGA-AD<sup>TM</sup> score (excluding subject's scalp)
- %BSA affected calculation (excluding subject's scalp)
- EASI (excluding subject's scalp)
- PP-NRS (by subject or caregiver)
- •

- AE recording
- Concomitant medication recording

#### 7.6 Unscheduled Visits

Unscheduled visits may occur, as needed. For subjects who experience suspected disease worsening (vIGA-AD<sup>TM</sup>  $\geq$  2) between scheduled study visits may contact the study site to arrange an unscheduled visit (see Section 5.1.5.2). The following assessments may be performed:

- Brief physical exam
- Vital signs measurements
- Urine pregnancy test (WOCBP)
- Blood sample collection for clinical laboratory tests (serum chemistry and hematology)
- Urinalysis
- vIGA-AD<sup>TM</sup> score (excluding subject's scalp)
- %BSA affected calculation (excluding subject's scalp)
- EASI (excluding subject's scalp)
- •
- PP-NRS (by subject or caregiver)
- AE recording
- Concomitant medication recording
- Collect and review subject diaries for treatment compliance, if applicable
- Dispense subject diaries, if applicable
- Collect and dispense study drug, if applicable
- Review instructions on how to apply study drug, if applicable
- Study drug application under supervision, if applicable

If disease worsening is confirmed, a new treatment course will be initiated.

## 7.7 Early Termination Visit

Subjects who withdraw early from the study will be asked to return to the study site to complete early termination assessments as follows:

- Brief physical examination
- Vital signs measurement
- Urine pregnancy test (WOCBP)
- Blood sample collection for clinical laboratory tests (serum chemistry and hematology)
- Urinalysis
- vIGA-AD<sup>TM</sup> score (excluding subject's scalp)
- %BSA affected calculation (excluding subject's scalp)
- EASI (excluding subject's scalp)

Protocol No.: DMVT-505-3103 Clinical Study Protocol



- AE recording
- Concomitant medication recording
- Collect subject diaries
- Review subject diaries for treatment compliance
- Collect study drug

# 7.8 End of Study

The end of study is defined as when the last active subject has completed the Week 49 Follow-up Visit one week after the end of treatment.

# 8 Safety Monitoring and Reporting

# 8.1 Adverse Events, Serious Adverse Events, and Adverse Events of Special Interest

The Investigator or site staff is responsible for detecting, documenting, and reporting events that meet the definition of an AE, SAE, or adverse event of special interest (AESI). At each visit/contact, subjects should be questioned in a general way so as not to introduce bias in detecting AEs and/or SAEs. Open-ended and non-leading verbal questioning of the subject is the preferred method to inquire about AE occurrence.

Investigators are not obligated to actively seek AEs or SAEs in former study subjects. However, if the Investigator learns of any SAE, including a death, at any time after a subject has been discharged from the study, and he/she considers the event reasonably related to the study drug or study participation, the Investigator should promptly notify the Sponsor.

A narrative will be written and included in the Clinical Study Report for all SAEs and AESIs, and for all AEs that lead to study discontinuation

#### **8.1.1** Definition of Adverse Events

An AE is any untoward medical occurrence in a subject temporally associated with the use of a medicinal product, whether considered causally related or not related to the medicinal product.

An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product.

Events meeting the definition of an AE include:

- Any abnormal laboratory test results (hematology, clinical chemistry) or other safety assessments (e.g., vital signs measurements), including those that worsen from Baseline, and felt to be clinically significant in the medical and scientific judgment of the Investigator
- Exacerbation of a chronic or intermittent pre-existing condition (e.g., plaque psoriasis) including either an increase in frequency and/or intensity of the condition
- For skin-related AEs, it should be noted whether or not the event is in the area of active application of study drug, and/or if spreading beyond the application site.
- New conditions detected or diagnosed after study drug administration even though it may have been present prior to the start of the study
- Signs, symptoms, or the clinical sequelae of a suspected interaction
- Signs, symptoms, or the clinical sequelae of a suspected overdose of either study drug or a concomitant medication (overdose per se will not be reported as an AE/SAE)
- "Lack of efficacy" or "failure of expected pharmacological action" per se will not be reported as an AE or SAE. Such instances will be captured in the efficacy assessments. However, the signs, symptoms, and/or clinical sequelae resulting from lack of efficacy will be reported as AE or SAE if they fulfill the definition of an AE or SAE.

Events that **do not** meet the definition of an AE include:

• Any clinically significant abnormal laboratory findings or other abnormal safety assessments that are associated with the underlying disease, unless judged by the Investigator to be more severe than expected for the subject's condition

- The disease/disorder being studied or expected progression, signs, or symptoms of the disease/disorder being studied, unless more severe than expected for the subject's condition
- Medical or surgical procedure (e.g., endoscopy, appendectomy); the condition that leads to the procedure is an AE


Clinical Study Protocol

- Situations where an untoward medical occurrence did not occur (social and/or convenience admission to a hospital)
- Anticipated day-to-day fluctuations of pre-existing disease(s) or condition(s) present or detected at the start of the study that do not worsen

#### 8.1.2 Definition of Serious Adverse Event

If an event is not an AE per Section 8.1.1, then it cannot be an SAE even if serious conditions are met (e.g., hospitalization for signs/symptoms of the disease under study, death due to progression of disease, etc.).

An SAE is any untoward medical occurrence that, at any dose:

- Results in death
- Is life-threatening
- The term "life threatening" refers to an event in which the subject was at risk of death at the time of the event. It does not refer to an event, which hypothetically might have caused death, if it were more severe.
- Requires hospitalization or prolongation of existing hospitalization
- In general, signifies that the subject has been detained (usually involving at least an overnight stay) at the hospital or emergency ward for observation and/or treatment that would not have been appropriate in the physician's office or outpatient setting. Complications that occur during hospitalization are AEs. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether "hospitalization" occurred or was necessary, the AE should be considered serious.
- Hospitalization for elective treatment of a pre-existing condition that did not worsen from Baseline is not considered an AE.
- Results in disability/incapacity: a substantial disruption of a person's ability to conduct normal life functions.
- This definition is not intended to include experiences of relatively minor medical significance such
  as uncomplicated headache, nausea, vomiting, diarrhea, influenza, and accidental trauma (e.g.,
  sprained ankle) which may interfere or prevent everyday life functions but do not constitute a
  substantial disruption.
- Results in a congenital anomaly/birth defect

Medical or scientific judgment should be exercised in deciding whether reporting is appropriate in other situations, such as important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the subject or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition. These should also be considered serious. Examples of such events are invasive or malignant cancers, intensive treatment in an emergency room or at home for

allergic bronchospasm, blood dyscrasias, or convulsions that do not result in hospitalization, or development of drug dependency or drug abuse.

# 8.1.3 Adverse Events of Special Interest

In prior clinical studies, contact dermatitis, folliculitis, and headache have been identified as AEs of particular clinical importance and will be reported as AESIs in this study whether or not the AE is considered related to study drug.

In each case study drug may be continued or discontinued, based on Investigator judgment, and may be restarted when the event resolves. In addition, the following information must be collected for each of these AESIs:

#### **Contact Dermatitis**

Contact dermatitis: the study site should collect location, duration, size, associated symptoms (itching, burning, pain), severity (mild, moderate, severe), time to onset, and photograph the affected site (if possible). If the subject or caregiver contacts the study site to report significant skin irritation at or near the site of study drug application between study visits, the subject should be brought in for an unscheduled visit, if possible.

#### Headache

The study site should collect duration, severity (mild, moderate, severe), time to onset, and location (e.g., frontal, temporal, occipital, diffuse).

#### **Follicular Event**

The study site should collect the location, duration, size, associated signs and symptoms (itching, burning, pain, erythema), severity (mild, moderate, severe), describe morphology [scale (keratotic/cornified) or no scale (non-keratotic/non-cornified)], time to onset, and photograph the affected site (if possible). Additional information regarding management of folliculitis is provided in Section 8.2.1.2.4.

In particular, the term 'folliculitis' may not correctly describe the morphology of the observed local follicular events as these appear to be more consistent with a keratoses pilaris-like follicular based papule. Tapinarof upregulates components of the stratum corneum, including involucrin, hornerin, and filaggrin and increased cornification at, and subsequent mechanical occlusion of, the follicular ostia has been suggested to be a potentially on target mechanism by which these lesions may develop in some individuals treated with tapinarof cream. Additional morphologic description will help to more fully and appropriately characterize these follicular events.

Possible descriptors include, but are not limited to:

- Folliculitis
  - Non-inflammatory
  - Inflammatory
- Milia
  - Non-inflammatory
  - Inflammatory
- Keratosis pilaris

Non-inflammatory

## - Inflammatory

Additional AESIs may be identified during the evaluation of safety data for the Clinical Study Report.

#### 8.2 Classification of Adverse Events

# 8.2.1 Assigning Severity Rating for Adverse Events

# 8.2.1.1 Criteria for Determining Adverse Event Severity

The Investigator will make an assessment of the severity of each AE and SAE according to the National Cancer Institute CTCAE, v. 5.0, 2017. For terms not specified with the CTCAE, the criteria in Table 5 should be used to determine the grade severity.

Table 5: Criteria for Determining the Grade/Severity of Adverse Event Terms Not Specified by the National Cancer Institute CTCAE

| Grade | Criteria |
|---|---|
| 1 | Mild; asymptomatic or mild symptoms, clinical or diagnostic observations only; intervention not indicated |
| 2 | Moderate; minimal, local, or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living <sup>a</sup> |
| 3 | Severe or medically significant but not immediately life threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living <sup>b</sup> |
| 4 | Life threatening consequences; urgent intervention indicated |
| 5 | Death related to adverse event |

a. Instrumental activities of daily living refer to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.

CTCAE = Common Terminology Criteria for Adverse Events.

AE severity should be recorded in the appropriate section of the AE CRF and in the subject's source documents.

#### 8.2.1.2 Toxicity Management Criteria

# 8.2.1.2.1 Grade 1 or Grade 2 Adverse Event

Subjects who develop a Grade 1 or Grade 2 AE may continue investigational product at the discretion of the Investigator. Subjects who choose to withdraw from study due to a Grade 1 or 2 AE should have study withdrawal/early termination evaluations completed.

#### 8.2.1.2.2 Grade 3 Adverse Event

Subjects who develop a Grade 3 AE should be managed as follows:

- If the Investigator has compelling evidence that the Grade 3 AE has not been caused by investigational product, then dosing may continue after discussion with the Medical Monitor.
- Subjects who develop a Grade 3 AE that the Investigator considers related to investigational
  product should have the investigational product discontinued. Subjects experiencing Grade 3 AEs
  requiring permanent discontinuation of investigational product should be followed weekly until
  resolution or stability of the AE and encouraged to have withdrawal study evaluations completed.

#### 8.2.1.2.3 Grade 4 Adverse Event

Subjects who develop a Grade 4 AE should have investigational product permanently discontinued.

b. Self-care activities of daily living refer to bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden.

Subjects experiencing Grade 4 AEs requiring permanent discontinuation of investigational product should be followed weekly until resolution or stability of the AE and encouraged to have withdrawal study evaluations completed.

#### 8.2.1.2.4 Folliculitis

Subjects using tapinarof topically may experience folliculitis. The majority of these events are mild or moderate and do not require intervention or interruption in study drug use. On close inspection, the morphology is similar to that of keratosis pilaris suggesting that the potential mechanism may be increased follicular cornification with subsequent follicular plugging. Importantly, AhR regulates the epidermal differentiation complex and tapinarof has been shown to repair the skin barrier through activation of stratum corneum components including fillagrin, hornerin and involucrin. This latter point suggests that the keratosis pilaris-like reaction may be an on-target effect predictive of a therapeutic response to tapinarof cream.

Several approaches can be employed to manage those patients with folliculitis who may be symptomatic including temporary interruption of study drug use at sites of folliculitis and/or the local application to affected areas of topical keratolytics such as 12% lactic acid lotion or 5-10% urea creams or lotions.

# 8.2.1.2.5 Other Management Criteria:

The Medical Monitor should be notified if any of the following occur:

• Severe signs or symptoms, or significant changes in any of the safety assessments, that put the safety of the subject at risk (e.g., laboratory tests or vital signs, etc.) as judged by the Investigator.

# 8.2.2 Assigning Causal Relationship to Study Drug

The Principal Investigator or sub-Investigator is to make the causality assessment. The reasonable possibility of the relationship of an AE to study drug is to be assessed with careful medical consideration at the time of evaluation of an AE. The following definitions are to be used for the relationship of the AE to study drug:

- Related: A clinical event, including laboratory test abnormality, with a temporal relationship to study drug administration that makes a causal relationship plausible, unlikely attributed to concurrent disease or other drugs or chemicals, and that follows a clinically reasonable response on re administration (rechallenge) or withdrawal (dechallenge), although information on drug withdrawal may be lacking or unclear.
- **Not related**: A clinical event, including laboratory test abnormality, with a temporal relationship to study drug administration that makes a causal relationship improbable and/or in which other drugs, chemicals, or underlying disease provide a plausible explanation.

Any AEs /SAEs assessed as related to study participation (e.g., protocol mandated procedures, invasive tests, or change in existing therapy) or related to study drug will be recorded from the time a subject consented to participate in the study up to and including any follow-up contact.

All AEs, whether related to study drug or not, must be fully and completely documented on the AE page of the CRF and in the subject's clinical record. In the event a subject is withdrawn from the study because of an AE, the primary reason for withdrawal (i.e., due to an AE) must be recorded on the CRF as such.

#### 8.3 Time Period and Frequency for Event Assessment and Follow-Up

# 8.3.1 Adverse Event Reporting

All AEs will be collected from the time of signed informed consent until the final visit.

Any AEs assessed as related to study participation (e.g., protocol mandated procedures, invasive tests, or change in existing therapy) will be collected from the time a subject consented to participate in the study up to and including any follow-up contact.

All SAEs will be recorded on the CRF and reported to the Sponsor within 24 hours via email or phone (refer to Medical Monitor / Sponsor Information Page for contact information) (see Section 8.4).

# 8.3.2 Follow-Up of Adverse Events

After the initial AE/SAE report, the Investigator is required to proactively follow each subject at subsequent visits/contacts. All SAEs and nonserious AEs will be followed until resolution, until the condition stabilizes, until the event is otherwise explained, or until the subject is lost to follow-up.

The Investigator will assess the outcome of each AE using the following criteria:

- Recovered/Resolved: The event has improved or subject recuperated.
- Recovered/Resolved with sequelae: The subject has recuperated but retained pathological conditions resulting from the prior disease or injury.
- **Recovering/Resolving:** The event is improving.
- Not recovered/Not resolved: The event has not improved or subject recuperated.
- Unknown: The outcome of the event is not known, not observed, not recorded, or refused.
- **Fatal:** Termination of life as an outcome of the AE.

# **8.4 Reporting Procedures**

# 8.4.1 Serious Adverse Event Reporting

When an Investigator determines that an AE meets the protocol definition of an SAE during the study, he/she must notify the Sponsor using an SAE Report Form within 24 hours of the study site personnel's knowledge of the event, regardless of the Investigator assessment of the relationship of the event to study drug. Relevant information will be entered on the AE page and on all other applicable pages of the CRF; source documentation should not be sent with the SAE Report Form unless requested.

Follow-up information received on SAEs should be emailed or faxed to the Sponsor within 1 business day of receipt (refer to Medical Monitor / Sponsor Information Page for contact information). This information should be included on a follow-up SAE form and filed with the original SAE information.

All SAEs will be followed until resolution, until the condition stabilizes, until the event is otherwise explained, or until the subject is lost to follow-up.

The completed SAE Report Form should be submitted via email or fax to the SAE Reporting Contact which can be found on the Medical Monitor / Sponsor Information Page of this protocol.

Do not delay reporting a suspected SAE in order to obtain additional information. Any additional information, if collected, can be reported as a follow-up to the initial report.

## 8.4.2 Regulatory Reporting Requirements for Serious Adverse Events

Prompt notification by the Investigator to the Sponsor of SAEs (even for non-interventional post-marketing studies) is essential so that legal obligations and ethical responsibilities towards the safety of subjects and the safety of a product under clinical investigation are met.

The Sponsor has a legal responsibility to notify both the local regulatory authority and other regulatory agencies about the safety of a product under clinical investigation. The Sponsor will comply with country-specific regulatory requirements relating to safety reporting to the regulatory authority, IRB/IEC, and investigators.

Investigator safety reports are prepared for suspected unexpected serious adverse reactions according to local regulatory requirements and are forwarded to Investigators as necessary.

An Investigator who receives an investigator safety report describing a SAE(s) or other specific safety information (e.g., summary or listing of SAEs) from the Sponsor will file it with the Investigator's Brochure and will notify the IRB/IEC, if appropriate, according to local requirements.

# 8.5 Pregnancy Management and Reporting

Any female subject who becomes pregnant during the study will be withdrawn. Details will be collected for all pregnancies in female subjects and female partners of male subjects that begin after the start of dosing and through the Follow-up visit. Pregnancy is not automatically considered an AE.

If a pregnancy is reported, then the Investigator should complete a Pregnancy Report Form and submit via email or fax to the Pregnancy Reporting Contact for which contact information can be found on the Medical Monitor / Sponsor Information Page of this protocol, within 2 weeks of learning of the pregnancy. The subject will also be followed to determine the outcome of the pregnancy. Information on the status of the mother and child will be forwarded to the Sponsor. Generally, follow-up will be no longer than 6 to 8 weeks following the estimated delivery date. Any premature termination of the pregnancy will be reported.

Any SAE occurring in association with a pregnancy brought to the Investigator's attention after the subject has completed the study and considered by the Investigator as possibly related to the study drug must be promptly reported to the Sponsor or the Sponsor's representative.

The Investigator must attempt to collect pregnancy information on any female partners of male study subjects who become pregnant while the subject is enrolled in the study. Pregnancy information must be reported to the Sponsor or the Sponsor's representative as described above. The partner will also be followed to determine the outcome of the pregnancy. Information on the status of the mother and child will be forwarded to Sponsor or the Sponsor's representative. Generally, follow-up will be no longer than 6 to 8 weeks following the estimated delivery date. Any premature termination of the pregnancy will be reported on the Pregnancy Report Form.

#### 9 Data Management

For this study, subject data will be entered into the Sponsor-defined CRFs, transmitted electronically to the Sponsor or designee, and combined with data provided from other sources in a validated data system.

Management of clinical data will be performed in accordance with applicable Sponsor standards and data cleaning procedures will be used to ensure the integrity of the data, e.g. errors will be corrected, and inconsistencies queried in the data.

Adverse events and relevant medical history will be coded using the most current version of the Medical Dictionary for Regulatory Activities. Concomitant medications will be coded with the most current version of World Health Organization Drug Global Dictionary.

The Investigator will retain original source documents and the Sponsor will receive CRF-required data as electronic datasets. Subject initials will not be collected or transmitted to the Sponsor.

## 10 Statistical Considerations and Data Analyses

This study is intended to show that tapinar fcream has a favorable safety and efficacy profile during repeated, intermittent treatment courses over an extended period of time.

#### 10.1 General Considerations

All study data will be summarized using descriptive statistics for the ITT population overall and by the following categories: received tapinarof treatment in either DMVT-505-3101 or DMVT-505-3102; received vehicle treatment in either DMVT-505-3101 or DMVT-505-3102; received tapinarof treatment in DMVT-505-2104; and enrolled directly into DMVT-505-3103. Categorical variables will be reported using frequency and percentage (e.g., sex, race). Continuous variables will be reported using number of subjects, mean, standard deviation (SD), median, minimum, and maximum. All efficacy and safety data will be listed by subject.

# 10.2 Determination of Sample Size

The sample size of this study is based on the ICH E1A guideline on extent of population exposure to assess clinical safety for drugs intended for long-term treatment of non-life-threatening conditions. Up to 961 subjects will be enrolled in this study across all regions, including up to 836 rollover subjects from studies DMVT-505-3101, DMVT-505-3102, and DMVT-505-2104 and approximately 125 subjects directly enrolling into this study.

#### **10.3 Analysis Populations**

All subjects enrolled into the study will be included in the ITT population.

# 10.4 Planned Analyses

All efficacy and safety measures over the course of the study will be presented. All analyses will be based on the ITT population. Details of planned analyses will be described in the Statistical Analysis Plan, which will be finalized prior to database lock.

#### 10.4.1 Disposition and Demographics

Demographic and baseline characteristics as well as medical history will be summarized using the ITT population, including frequency and percentages for categorical variables and mean, SD, median, minimum, and maximum for continuous variables.

The numbers of subjects will be summarized by the following categories: received tapinarof treatment in either DMVT-505-3101 or DMVT-505-3102; received vehicle treatment in either DMVT-505-3101 or DMVT-505-3102; received tapinarof treatment in DMVT-505-2104; and enrolled directly into DMVT-505-3103.

# **10.4.2 Efficacy Analyses**

All efficacy analyses will be performed based on the ITT population as described above. Summaries will be presented overall and by the following categories: received tapinarof treatment in either DMVT-505-3101 or DMVT-505-3102; received vehicle treatment in either DMVT-505-3101 or DMVT-505-3102; received tapinarof treatment in DMVT-505-2104; and enrolled directly into DMVT-505-3103. Summaries of efficacy endpoints by visit will be performed using OC and LOCF methods.

Efficacy endpoints are as follows:

For subjects entering the study with a vIGA-AD<sup>TM</sup> score of clear (0):

•

• Proportion of subjects who never experience vIGA-AD<sup>TM</sup>  $\geq 2$  throughout the study


Clinical Study Protocol

For subjects entering the study with a vIGA-AD<sup>TM</sup> score  $\geq 2$ :

• Proportion of subjects who achieve vIGA-AD<sup>TM</sup> = 0 or 1 at least 1 time during the study

The following endpoints will be summarized over subjects in the ITT population:

•

• change and percent change from Baseline in %BSA affected by visit (OC and LOCF)

LOCF)

• change and percent change from Baseline in EASI score by visit (OC and LOCF)

 Proportion of subjects with ≥ 50% improvement in EASI score from Baseline by visit (OC and LOCF)

 Proportion of subjects with ≥ 75% improvement in EASI score from Baseline by visit (OC and LOCF)

 Proportion of subjects with ≥ 90% improvement in EASI score from Baseline by visit (OC and LOCF)

• Mean change in PP- NRS score from Baseline at each study visit

• Proportion of subjects with a Baseline PP-NRS score ≥ 4 who achieve ≥ 4-point reduction in the PP-NRS from Baseline at each study visit




For analyses of time to event, such as the time to first worsening (vIGA-AD<sup>TM</sup>  $\geq$  2) or the time to first reaching a vIGA-AD<sup>TM</sup> score of 0, the Kaplan-Meier product limit method will be used to estimate the median time (if estimable). If the median is not estimable (e.g., < 50% of subjects reach the event), other methods for estimating the median and/or other percentiles will be applied.

The remaining efficacy endpoints will be summarized descriptively as follows: continuous data will include the mean, SD, minimum, maximum, median, and number of observations; descriptive summary statistics for categorical data will include frequency counts and percentages.

# **10.4.3 Safety Analyses**

The ITT Population will be used in the analysis of safety data. Summaries will be presented overall and by the following categories: received tapinarof treatment in either DMVT-505-3101 or DMVT-505-3102; received vehicle treatment in either DMVT-505-3101 or DMVT-505-3102; received tapinarof treatment in DMVT-505-2104; and enrolled directly into DMVT-505-3103.

The number and percent of subjects with TEAEs will be summarized by system organ class, and preferred term for all TEAEs, all TEAEs considered by the Investigator to be related to study drug, all SAEs, all TEAEs leading to study drug discontinuation, and all TEAEs leading to study discontinuation. TEAEs will be defined as follows:

- For rollover subjects, all AEs reported in DMVT-505-3103 will be considered to be a TEAE except for those AEs ongoing at the end of the parent study (DMVT-505-3101, DMVT-505-3102, or DMVT-505-2104) but resolved prior to the Visit 1 date in DMVT-505-3103.
- For subjects enrolled directly into DMVT-505-3103, all AEs that start after the first dose of study medication will be considered to be a TEAE.

Data listings will be provided for subjects who discontinued the study due to an AE and for subjects with an SAE.

Laboratory values will be classified as normal, low or high based on normal ranges supplied by the laboratory. Changes from Baseline in abnormality status will be summarized using shift tables. For quantitative laboratory measures, observed values and changes from Baseline will be summarized descriptively by visit.

Observed vital sign values (systolic and diastolic blood pressure, pulse rate, and body temperature) and change from Baseline in vital signs will be summarized similarly to the laboratory values.

LTS scores will be summarized by visit for subject (or caregiver) overall assessment and Investigator overall assessment separately.



Protocol No.: DMVT-505-3103 Clinical Study Protocol



# 10.5 Interim Analyses

A data-cut will be made at the time of preparation of the marketing application to present interim results; the final analysis will be conducted after study completion (e.g., the last subject's last visit).

# 10.6 Handling of Missing Data

Summaries of efficacy endpoints by visit will be performed using OC and LOCF methods.

# 11 Responsibilities

# 11.1 Investigator Responsibilities

#### 11.1.1 Good Clinical Practice

The Investigator will ensure that this study is conducted in accordance with the principles of the "Declaration of Helsinki" (as amended in Edinburgh, Tokyo, Venice, Hong Kong, and South Africa), ICH guidelines, or with the laws and regulations of the country in which the research is conducted, whichever affords the greater protection to the study subject. For studies conducted under a United States Investigational New Drug Application, the Investigator will ensure that the basic principles of "Good Clinical Practice," as outlined in 21 Code of Federal Regulations (CFR) 312, subpart D, "Responsibilities of Sponsors and Investigators," 21 CFR, part 50, 1998, and 21 CFR, part 56, 1998, are adhered to. These standards are consistent with the requirements of the European Community Directive 2001/20/EC.

Since this is a "covered" clinical trial, the Investigator will ensure that 21 CFR, Part 54, 1998, is adhered to; a "covered" clinical trial is any "study of a drug or device in humans submitted in a marketing application or reclassification petition subject to this part that the applicant or Food and Drug Administration relies on to establish that the product is effective (including studies that show equivalence to an effective product) or that make a significant contribution to the demonstration of safety." This requires that Investigators and all sub-Investigators must provide documentation of their financial interest or arrangements with the Sponsor, or proprietary interests in the drug being studied. This documentation must be provided before participation of the Investigator and any sub-Investigator. The Investigator and sub-Investigator agree to notify the Sponsor of any change reportable interests during the study and for 1 year following completion of the study. Study completion is defined as the date that the last subject has completed the protocol-defined activities.

# 11.1.2 Institutional Review Board/Independent Ethics Committee Approval

This protocol and any accompanying material to be provided to the subject (such as advertisements, subject information sheets, or descriptions of the study used to obtain informed consent) will be submitted by the Investigator or on behalf of the Investigator to an IRB or IEC. Approval from the IRB or IEC must be obtained before starting the study and should be documented in a letter to the Investigator specifying the protocol number, protocol version, protocol date, documents reviewed, and date on which the committee met and granted the approval.

Any modifications made to the protocol after receipt of IRB or IEC approval must also be submitted to the IRB or IEC for approval before implementation.

## 11.1.3 Informed Consent/Assent

The Investigator is responsible for obtaining written informed consent/assent from each individual participating in this study after adequate explanation of the aims, methods, objectives, and potential hazards of the study and before undertaking any study-related procedures. The Investigator must utilize an IRB- or IEC-approved consent form for documenting written informed consent. Each informed consent/assent will be appropriately signed and dated by the subject or the subject's legally authorized representative and the person obtaining consent.

#### 11.1.4 Confidentiality

The Investigator must assure that subjects' anonymity will be strictly maintained and that their identities are protected from unauthorized parties. Only subject number, date of birth, and an identification code (i.e., not

names) should be recorded on any form or biological sample submitted to the Sponsor, IRB or IEC, or laboratory. The Investigator must keep a log showing codes, names, and addresses for all subjects enrolled in the trial.

The Investigator agrees that all information received from the Sponsor, including but not limited to the Investigator Brochure, this protocol, CRFs, the investigational new drug, and any other study information, remain the sole and exclusive property of the Sponsor during the conduct of the study and thereafter. This information is not to be disclosed to any third party (except employees or agents directly involved in the conduct of the study or as required by law) without prior written consent from the Sponsor. The Investigator further agrees to take all reasonable precautions to prevent the disclosure by any employee or agent of the study site to any third party or otherwise into the public domain.

# 11.1.5 Study Files and Retention of Records

The Investigator must maintain adequate and accurate records to enable the conduct of the study to be fully documented and the study data to be subsequently verified. These documents should be classified into at least the following 2 categories: (1) Investigator's study file, and (2) subject clinical source documents.

The Investigator's study file will contain the protocol/amendments, CRF and query forms, IRB or IEC and governmental approval with correspondence, informed consent, drug records, staff curriculum vitae and authorization forms, and other appropriate documents and correspondence.

The required source data should include at least the following information for each subject:

- Subject identification (name, date of birth, gender)
- Documentation that subject meets eligibility criteria, i.e., history, physical examination, and confirmation of diagnosis (to support inclusion and exclusion criteria)
- Participation in trial (including trial number)
- Trial discussed and date of informed consent
- Dates of all visits
- Documentation that protocol-specific procedures were performed
- Results of efficacy parameters, as required by the protocol
- Start and end dates (including dose regimen) of trial medication (preferably drug dispensing and return should be documented as well)
- Record of all adverse events and other safety parameters (start and end date, and preferably including causality and intensity)
- Concomitant medication (including start and end dates, dose if relevant; dose changes should be recorded)
- Date of trial completion and reason for early discontinuation, if applicable

All clinical study documents must be retained by the Investigator until at least 2 years after the last approval of a marketing application in an ICH region (i.e., United States, Europe, or Japan) and until there are no pending or contemplated marketing applications in an ICH region; or, if no application is filed or if the application is not approved for such indication, until 2 years after the investigation is discontinued and regulatory authorities have been notified. Investigators may be required to retain documents longer if

required by applicable regulatory requirements, by local regulations, or by an agreement with the Sponsor. The Investigator must notify the Sponsor before destroying any clinical study records.

Should the Investigator wish to assign the study records to another party or move them to another location, the Sponsor must be notified in advance.

If the Investigator cannot guarantee this archiving requirement at the study site for any or all of the documents, special arrangements must be made between the Investigator and the Sponsor to store these in sealed containers outside of the site so that they can be returned sealed to the Investigator in case of a regulatory audit. When source documents are required for the continued care of the subject, appropriate copies should be made for storage outside of the site.

# 11.1.6 Electronic Case Report Forms

For each subject enrolled, a CRF must be completed and signed by the Investigator. This also applies to records for those subjects who fail to complete the study. If a subject withdraws from the study, the reason must be noted on the CRF. If a subject is withdrawn from the study because of a treatment-limiting AE, thorough efforts should be made to clearly document the outcome.

# 11.1.7 Drug Accountability

The Investigator or designee (i.e., pharmacist) is responsible for ensuring adequate accountability of all used and unused investigational medicinal product. This includes acknowledgment of receipt of each shipment of study product (quantity and condition), subject dispensing records, and returned or destroyed study product. Dispensing records will document quantities received from the Sponsor and quantities dispensed to subjects, including kit or lot number, date dispensed, subject identifier number, and the initials of the person dispensing the medication.

At study initiation, the monitor will evaluate the site's procedure for investigational medicinal product disposal/destruction in order to ensure that it complies with the Sponsor requirements. At the end of the study, following final drug inventory reconciliation by the monitor, the study site will dispose of and/or destroy all unused investigational medicinal product supplies, including empty containers, according to these procedures. If the site cannot meet the Sponsor's requirements for disposal, arrangements will be made between the site and the Sponsor or its representative for destruction or return of unused investigational medicinal product supplies.

All drug supplies and associated documentation will be periodically reviewed and verified by the study monitor over the course of the study.

## 11.1.8 Inspections

The Investigator should understand that source documents for this trial should be made available to appropriately qualified personnel from the Sponsor or its representatives, to IRBs or IECs, or to regulatory authority or health authority inspectors.

# 11.1.9 Protocol Compliance

The Investigator is responsible for ensuring the study is conducted in accordance with the procedures and evaluations described in this protocol.
## 11.2 Sponsor Responsibilities

## 11.2.1 Protocol Modifications

Protocol modifications, except those intended to reduce immediate risk to study subjects, may be made only by the Sponsor. All protocol modifications must be submitted to the IRB or IEC and regulatory authorities in accordance with local requirements. Approval must be obtained before changes can be implemented.

# 11.2.2 Study Report and Publications

A clinical study report will be prepared and provided to the regulatory agency(ies). The Sponsor will ensure that the report meets the standards set out in the ICH Guideline for Structure and Content of Clinical Study Reports (ICH E3). Note that an abbreviated report may be prepared in certain cases.

After conclusion of the study and without prior written approval from Dermavant Sciences, Inc., Investigators in this study may communicate, orally present, or publish in scientific journals or other scholarly media only after the following conditions have been met:

- The results of the study in their entirety have been publicly disclosed by or with the consent of Dermavant Sciences, Inc., in an abstract, manuscript, or presentation form; OR
- The study has been completed at all study sites for at least 5 years.

No such communication, presentation, or publication will include Dermavant Sciences, Inc. confidential information (see Section 11.1.4).

The Investigator will submit any proposed publication or presentation along with the respective scientific journal or presentation forum at least 30 days before submission of the publication or presentation. The Investigator will comply with Dermavant Sciences, Inc. request to delete references to its confidential information (other than the study results) in any paper or presentation and agrees to withhold publication or presentation for an additional 60 days in order to obtain patent protection if deemed necessary.

## 11.2.3 Posting of Information on Publicly Available Clinical Trial Registers

Study information from this protocol will be posted on publicly available clinical trial registers as required by applicable regulations. Results will be posted as required.

# 11.3 Joint Investigator/Sponsor Responsibilities

### 11.3.1 Access to Information for Monitoring

In accordance with ICH Good Clinical Practice guidelines, the study monitor must have direct access to the Investigator's source documentation in order to verify the data recorded in the CRFs for consistency.

The monitor is responsible for routine review of the CRFs at regular intervals throughout the study to verify adherence to the protocol and the completeness, consistency, and accuracy of the data being entered on them. The monitor should have access to any subject records needed to verify the entries on the CRFs. The Investigator agrees to cooperate with the monitor to ensure that any problems detected in the course of these monitoring visits are resolved.

In the event of COVID-19-like situation necessitating a limit on in-person contact, remote monitoring may be performed.

## 11.3.2 Access to Information for Auditing or Inspections

To ensure compliance with Good Clinical Practices and all applicable regulatory requirements, Dermavant Sciences, Inc. may conduct a quality assurance audit.


Clinical Study Protocol

Authorized representatives of Dermavant Sciences, Inc., a regulatory authority, an Independent Ethics Committee or an Institutional Review Board may visit the site to perform audits or inspections, including source data verification. The purpose of a Dermavant Sciences, Inc. audit or inspection is to systematically and independently examine all study-related activities and documents to determine whether these activities were conducted, and data were recorded, analyzed, and accurately reported according to the protocol, Good Clinical Practice guidelines of the ICH, and any applicable regulatory requirements. The Investigator should contact Dermavant Sciences, Inc. immediately if contacted by a regulatory agency about an inspection.

Representatives of regulatory authorities or of the Sponsor may conduct inspections or audits of the clinical study. If the Investigator is notified of an inspection by a regulatory authority the Investigator agrees to notify the Sponsor Medical Monitor immediately. The Investigator agrees to provide to representatives of a regulatory agency or the Sponsor access to records, facilities, and personnel for the effective conduct of any inspection or audit.

# 11.3.3 Study Discontinuation

The Sponsor reserves the right to terminate the study at any time. Should this be necessary, the Sponsor will arrange discontinuation procedures and notify the appropriate regulatory authority(ies), IRBs, and IECs. In terminating the study, the Sponsor and the Investigator will assure that adequate consideration is given to the protection of the subjects' interests.

#### 12 References

Bieber T. Atopic dermatitis. N Engl J Med. 2008 Apr 3;358(14):1483-94.

Cappon GD and Hurtt ME. Developmental toxicity of the kidney. In: Kapp RW and Yyl L, editors. Reproductive Toxicology, Target Organ Series, 3rd edition. New York:Informa Healthcare, 2010:193-204.

Carroll CL, Balkrishnan R, Feldman SR, Fleischer AB Jr, Manual JC. The burden of atopic dermatitis: impact on the patient, family, and society. Pediatr Dermatol. 2005; 22: 192-9.


Clinical Study Protocol

Frazier KS and Seely JC. Urinary system. In: Sahota PS, Popp JA, Hardisty JF and Gopinath C, editors. Toxicologic Pathology: Nonclinical Safety Assessment. CRC Press, 2013:421-84.

Furue M., Hashimoto-Hachiya A., Tsuji G. Aryl Hydrocarbon Receptor in Atopic Dermatitis and Psoriasis. Int J Mol Sci. 2019; 20: 5424.

Hanifin JM, Rajka G. Diagnostic features of atopic dermatitis. Acta Dermato-Venereologica Supplementum. 1980;92:44-7.

Hanifin JM, Thurston M, Omoto M, Cherill R, Tofte SJ, Graeber M. The eczema area and severity (EASI) index: assessment of reliability in atopic dermatitis. Experimental Dermatol. 2001: 10:11-18.

Lewis-Jones S. quality of life and childhood atopic dermatitis: the misery of living with childhood eczema, In J Clin Pract. 2006; 60:984-92.

Smith SH, Jayawickreme C, Rickard DJ, Nicodeme E, Bui T, Simmons C, Coquery CM, Neil J, Pryor WM, Mayhew D, Rajpal DK, Creech K, Furst S, Lee J, Wu D, Rastinejad F, Willson TM, Viviani F, Morris DC, Moore JT, Cote-Sierra J. Tapinarof Is a Natural AhR Agonist that Resolves Skin Inflammation in Mice and Humans. Journal of Invest Dermatol. 2017; 137: 2110–2119.

Zoetis T and Hurtt ME. Species comparison of anatomical and functional renal development. Birth Defects Research Part B. 2003;68:111-120.

## 13 Appendices

# Appendix 1. Hanifin and Rajka Criteria for Atopic Dermatitis Diagnosis

Major Criteria (must have at least three)

- Pruritus
- Typical morphology and distribution:
- Adults: flexural lichenification or linearity
- Children and infants: involvement of facial and extensor surfaces
- Chronic or chronically relapsing dermatitis
- Personal or family history of atopy (asthma, allergic rhinitis, atopic dermatitis)

Minor Criteria (must have at least three)

- Xerosis
- Ichthyosis/keratosis pilaris/palmar hyperlinearity
- Immediate (Type 1) skin test reactivity
- Elevated serum IgE
- Early age at onset
- Tendency to skin infections (Staphylococcus aureus, herpes simplex)/impaired cellular immunity
- Tendency to nonspecific hand/foot dermatitis
- Nipple eczema
- Cheilitis
- Recurrent conjunctivitis
- Dennie-Morgan infraorbital fold
- Keratoconus
- Anterior subcapsular cataracts
- Orbital darkening
- Facial pallor/erythema
- Pityriasis alba
- Anterior neck folds
- Itch when sweating
- Intolerance to wool and lipid solvents
- Perifollicular accentuation
- Food intolerance
- Course influenced by environmental/emotional factors
- White dermographism/delayed blanch

Source: Hanifin, 1980.

# **Appendix 2. Fitzpatrick Skin Type Scale**

| Skin Type | Sunburn Tendency | Suntan Tendency |
|-----------|---------------------|-----------------|
| Type I | Always burns easily | Never tan |
| Type II | Always burns easily | Tans slightly |
| Type III | Burns moderately | Tans gradually |
| Type IV | Burns minimally | Tans moderately |
| Type V | Rarely burns | Tans profusely |
| Type VI | Never burns | Tans profusely |


Clinical Study Protocol

# Appendix 5. Validated Investigator Global Assessment Scale for Atopic Dermatitis

## **Instructions:**

The vIGA-AD<sup>TM</sup> score is selected using the descriptors below that best describe the overall appearance of the lesions (excluding lesions on the scalp) at a given time point. It is not necessary that all characteristics under Morphological Description be present.


Clinical Study Protocol

| Score | Morphological Description |
|---|---|
| 0 – Clear | No inflammatory signs of atopic dermatitis (no erythema, no induration/papulation, no lichenification, no oozing/crusting). Post-inflammatory hyperpigmentation and/or hypopigmentation may be present. |
| 1 – Almost clear | Barely perceptible erythema, barely perceptible induration/papulation, and/or minimal lichenification. No oozing or crusting. |
| 2 – Mild | Slight but definite erythema (pink), slight but definite induration/papulation, and/or slight but definite lichenification. No oozing or crusting. |
| 3 – Moderate | Clearly perceptible erythema (dull red), clearly perceptible induration/papulation, and/or clearly perceptible lichenification. Oozing and crusting may be present. |
| 4 – Severe | Marked erythema (deep or bright red), marked induration/papulation, and/or marked lichenification. Disease is widespread in extent. Oozing or crusting may be present. |

### **Notes:**

1. In indeterminate cases, please use extent to differentiate between scores.

# For example:

Patient with marked erythema (deep or bright red), marked papulation and/or marked lichenification that is limited in extent, will be considered "3 – Moderate".

2. Excoriations should not be considered when assessing disease severity.

Copyright ©2017 Eli Lilly and Company – Used with the permission of Eli Lilly and Company under a Creative Commons Attribution-No Derivatives 4.0 International License – https://creativecommons.org/licenses/by-nd/4.0/.

# Appendix 6. Calculation of Percent Body Surface Area Affected and Eczema Area Severity Index Calculation of %BSA Affected

NOTE: At Baseline and for all efficacy assessments, lesions on the scalp will not be included in the calculation of %BSA affected as these areas will not be included in the efficacy analyses.

Measurement of involved BSA is estimated by the handprint method: the total palmar surface of the subject's palm and digits is approximately 1% of their total BSA.

Estimate the involved regional area by determining the number of "full" handprints plus the number of handprints covered if several smaller lesions are "pushed together."

For subjects ages 8 years and above the maximum involvement by region is as follows:

- Head and neck = 10% of overall BSA (10 handprints);
   1 hand-sized lesion ~ 10% of head and neck area
- Arms/Upper extremities = 20% of overall BSA (20 handprints);
   1 hand-sized lesion ~ 5% of the upper extremities
- Trunk (including axillae and groin) = 30% of overall BSA (30 handprints);
   1 hand-sized lesion ~ 3.33% of the trunk
- Legs/Lower extremities (including buttocks) = 40% of overall BSA (40 handprints); 1 hand-sized lesion  $\sim 2.5\%$  of the lower extremities

For subjects ages <8 years the maximum involvement by region is as follows:

- Head and neck = 20% of overall BSA (20 handprints);
   1 hand-sized lesion ~ 5% of head and neck area
- Arms/Upper extremities = 20% of overall BSA (20 handprints);
   1 hand-sized lesion ~ 5% of the upper extremities
- Trunk (including axillae and groin) = 30% of overall BSA (30 handprints); 1 hand-sized lesion ~ 3.33% of the trunk
- Legs/Lower extremities (including buttocks) = 30% of overall BSA (30 handprints); 1 hand-sized lesion ~ 3.33% of the lower extremities

Table 6: Calculation of Percent Body Surface Area Affected

| Body Region | Number of Handprints for<br>Each Region |
|---|---|
| Head and neck | |
| Arms/upper extremities | |
| Trunk | |
| Legs/lower extremities | |
| TOTAL Involved %BSA – sum of handprints for each region | |

Note: Shaded cells will be calculated in the CRF.

%BSA = percent body surface area; CRF = case report form

## **Calculation of EASI score (scalp excluded)**

Four anatomic sites – head, upper extremities, trunk, and lower extremities – are assessed for erythema, edema/papulation, excoriation and lichenification as seen on the day of the examination. The severity of each sign is assessed using a 4-point scale, half points may be used (e.g. 0.5, 1.5, 2.5):


Clinical Study Protocol

0 = Absent

1 = Mild

2 = Moderate

3 = Severe

The area affected by AD within a given anatomic site is estimated as a percentage of the total area of that anatomic site, based on the %BSA calculation, and assigned a numerical value according to the degree of AD involvement. For the purpose of assigning a numerical value for each anatomic site, %BSA ranges will be used as follows:

0 = no (0%) involvement

1 = > 0% to < 9.50% involvement

 $2 = \ge 9.50\%$  to < 29.50% involvement

 $3 = \ge 29.50\%$  to < 49.50% involvement

 $4 = \ge 49.50\%$  to < 69.50% involvement

5 = 89.50% to 89.50% involvement

 $6 = \ge 89.50\%$  to 100% involvement

The EASI score will be calculated in the CRF based on the subject's age, the rating scores for each region, and the number of handprints involved for each region.

Table 7: Calculation of Eczema Area and Severity Index Score for Ages 8 Years and Above


Clinical Study Protocol

| Characteristic of lesions | Rating Score | | Body 1 | region | |
|---|---|---|---|---|---|
| | | Head and Neck | Arms / Upper<br>Extremities | Trunk | Legs / Lower<br>Extremities |
| Erythema | 0 = None (Absent) | | | | |
| Edema/Papulation | 1 = Mild | | | | |
| Lichenification | 2 = Moderate | | | | |
| Excoriation | 3 = Severe | | | | |
| Add together each of the 4 s | cores for each of the bo | dy regions to give 4 s | separate subtotals | | |
| Subtotals | | A1 = | A2 = | A3 = | A4 = |
| From the BSA calculation in percentage into a value from | | dy region using the F | Regional %BSA Inv | volvement column t | to covert that |
| Number of Handprints | | | | | |
| Multiplier for body region | | 10 | 5 | 3.33 | 2.5 |
| Percentage for each Region | | % | % | % | % |
| Area of involvement for<br>each body region affected<br>Score between 0 and 6 for<br>each region | 0 = 0%<br>1 = 1-9%<br>2 = 10-29%<br>3 = 30-49%<br>4 = 50-69%<br>5 = 70-89%<br>6 = 90-100% | | | | |
| | | B1 = | B2 = | B3 = | B4 = |
| For each body region, multiplier to give 4 subtotals | | , and A4 by the degree | ee of body involven | nent (B1, B2, B3, an | nd B4) and |
| | | C1 = A1 x B1 x<br>0.1 | C2 = A2 x B2 x<br>0.2 | C3 = A3 x B3 x<br>0.3 | C4 = A4 x B4 x<br>0.4 |
| | | C1 = | C2 = | C3 = | C4 = |
| The subject's EASI score is | the sum of C1+C2+C3- | +C4 | | EASI = | |

Hanifin JM et al. Copyright © 2001 Munksgaard. Reproduced with permission of Blackwell Publishing Ltd
Note: Shaded cells are either fixed values or will be calculated in the CRF. Multiplier is a fixed number representing fraction of
total body area. The number of handprints will be imputed from data entered for the calculation of %BSA affected.
%BSA = percent body surface area; BSA = body surface area; CRF = case report form; EASI = Eczema Area and Severity Index

Calculation of Eczema Area and Severity Index Score for Ages < 8 Years Table 8:

| Characteristic of lesions | Rating Score | | Body 1 | region | |
|---|---|---|---|---|---|
| | | Head and Neck | Arms / Upper<br>Extremities | Trunk | Legs / Lower<br>Extremities |
| Erythema | 0 = None (Absent) | | | | |
| Edema/Papulation | 1 = Mild | | | | |
| Lichenification | 2 = Moderate | | | | |
| Excoriation | 3 = Severe | | | | |
| Add together each of the 4 so | cores for each of the bo | dy regions to give 4 s | eparate subtotals | | |
| Subtotals | | A1 = | A2 = | A3 = | A4 = |
| From the BSA calculation in percentage into a value from | | dy region using the R | legional %BSA Inv | volvement column t | o covert that |
| Number of Handprints | | | | | |
| Multiplier for body region | | 5 | 5 | 3.33 | 3.33 |
| Percentage for each Region | | % | % | % | % |
| Area of involvement for | 0 = 0% | | | | |
| each body region affected | 1 = 1-9% | | | | |
| Score between 0 and 6 for | 2 = 10-29% | | | | |
| each region | 3 = 30-49% | | | | |
| | 4 = 50-69% | | | | |
| | 5 = 70-89% | | | | |
| | 6 = 90-100% | | | | |
| | | B1 = | B2 = | B3 = | B4 = |
| For each body region, multip<br>multiplier to give 4 subtotals | | , and A4 by the degre | ee of body involven | nent (B1, B2, B3, ar | nd B4) and |
| | | $C1 = A1 \times B1 \times$ | $C2 = A2 \times B2 \times$ | $C3 = A3 \times B3 \times$ | $C4 = A4 \times B4 \times$ |
| | | 0.2 | 0.2 | 0.3 | 0.3 |
| | | C1 = | C2 = | C3 = | C4 = |
| The subject's EASI score is | the sum of C1+C2+C3- | +C4 | | EASI = | |

Clinical Study Protocol

Hanifin JM et al. Copyright © 2001 Munksgaard. Reproduced with permission of Blackwell Publishing Ltd Note: Shaded cells are either fixed values or will be calculated in the CRF. Multiplier is a fixed number representing fraction of total body area. The number of handprints will be imputed from data entered for the calculation of %BSA affected. %BSA = percent body surface area; BSA = body surface area; CRF = case report form; EASI = Eczema Area and Severity Index

The EASI score is obtained by using one of the below formulas, based on the subject's age:

For children age 8 years and older:

EASI = 
$$0.1 (E_h + I_h + Ex_h + L_h) A_h + 0.2 (E_u + I_u + Ex_u + L_u) A_u + 0.3 (E_t + I_t + Ex_t + L_t) A_t + 0.4 (E_l + I_l + Ex_l + L_l) A_l$$

For children under the age of 8 years:

EASI = 0.2 
$$(E_h + I_h + Ex_h + L_h)$$
 A<sub>h</sub> + 0.2  $(E_u + I_u + Ex_u + L_u)$  A<sub>u</sub> + 0.3  $(E_t + I_t + Ex_t + L_t)$  A<sub>t</sub> + 0.3  $(E_l + I_l + Ex_l + L_l)$  A<sub>l</sub>

Where E, I, Ex, L and A denote erythema, induration, excoriation, lichenification and area, respectively, and h, u, t, and l denote head, upper extremities, trunk, and lower extremities, respectively.

# Appendix 7. Summary Table of Patient Reported Outcomes and Quality of Life Assessments Completed by Age

| Subject's Age<br>at Time of<br>Consent <sup>a</sup> | | PP-NRS |
|---|---|---|
| 2 | | PP-NRS |
| | | (Caregiver) |
| 3 | | PP-NRS |
| | | (Caregiver)<br>PP-NRS |
| 4 | | (Caregiver) |
| | | PP-NRS |
| 5 | | (Caregiver) |
| | - | PP-NRS |
| 6 | | (Caregiver) |
| | | PP-NRS |
| 7 | | (Caregiver) |
| | | PP-NRS |
| 8 | | (Caregiver) |
| | - | PP-NRS |
| 9 | | (Caregiver) |
| | | PP-NRS |
| 10 | | (Caregiver) |
| | | PP-NRS |
| 11 | | (Caregiver) |
| | | PP-NRS |
| 12 | | (Subject) |
| 10 | | PP-NRS |
| 13 | | (Subject) |
| 1.4 | | PP-NRS |
| 14 | | (Subject) |
| 1.5 | | PP-NRS |
| 15 | | (Subject) |
| 1.0 | | PP-NRS |
| 16 | | (Subject) |
| 1.7 | | PP-NRS |
| 17 | | (Subject) |
| 101 | | PP-NRS |
| 18+ | | (Subject) |

a. For rollover subje mined as age at the time of consent in the parent study. For direct-enrolling subjects, age is determined as age at the time of consent in this study. In both cases, the determined age will remain the same throughout the duration of this study for the purposes of completing all assessments.

PP-NRS = Peak Pruritus Numeric

Rating Scale.

# **Appendix 13. Peak Pruritus-Numeric Rating Scale**

The PP-NRS is a scale used to quickly assess itch/pruritus severity over a 24-hour period which will be used daily to assess peak pruritus.


Clinical Study Protocol

For subjects ages 2 to < 12 years, the PP-NRS will be completed by the caregiver. For subjects ages  $\geq$  12 years, the PP-NRS will be completed by the subject.

# **PP-NRS**

On a scale of 0 to 10, with 0 being 'no itch' and 10 being 'worst itch imaginable', how would you rate your itch at the worst moment during the previous 24 hours?



PP-NRS © 2019 Regeneron Pharmaceuticals, Inc. and SAR&D. All rights reserved. Used with permission of Regeneron Pharmaceuticals, Inc. and SAR&D

Clinical Study Protocol